

## CLINICAL STUDY PROTOCOL

Study Title: A Phase 3b, Multicenter, Open-Label Study to Investigate the Efficacy

and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination in Treatment-Naïve and Treatment-Experienced Subjects with Chronic

Genotype 1 HCV Infection

**Sponsor:** Gilead Sciences, Inc.

333 Lakeside Drive

Foster City, CA 94404, USA

IND Number: Not Applicable EudraCT Number: Not Applicable

Clinical Trials.gov

Identifier: NCT02021656

**Indication:** Hepatitis C Virus Infection

Protocol ID: GS-US-337-0131

Gilead Study Director: Name: Jenny Yang, PharmD

Telephone: PPD Fax: PPD E-mail: PPD

Protocol Version/Date: Original: 28 May 2013

Amendment 1.1: 12 December 2013 Amendment 2.0: 01 August 2014 Amendment 3.0: 12 February 2016

#### CONFIDENTIALITY STATEMENT

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# **TABLE OF CONTENTS**

| TA | BLE OF | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF I | N-TEXT TABLES | 4 |
| PRO | ЭТОСС | OL SYNOPSIS | 5 |
| GL | OSSAR | Y OF ABBREVIATIONS AND DEFINITION OF TERMS | 12 |
| 1. | INTR | ODUCTION | 16 |
| | 1.1. | Background | |
| | 1.1. | 1.1.1. HCV Infection | |
| | | 1.1.2. HCV Infection in Korea | |
| | | 1.1.3. HCV Infection in Taiwan | |
| | | 1.1.4. HCV Infection in China | |
| | | 1.1.5. Summary | |
| | 1.2. | Sofosbuvir (formerly GS-7977) and Ledipasvir (formerly, GS-5885) Fixed Dose Combination | 20 |
| | | 1.2.1. General Information | 20 |
| | | 1.2.2. Summary of Additional Clinical Experience with Sofosbuvir and Ledipasvir | 21 |
| | 1.3. | Rationale for This Study | |
| | 1.4. | Rationale for Dose Selection of SOF/LDV FDC | |
| | 1.5. | Overall Risk/Benefit Assessment | |
| | 1.6. | Compliance | |
| 2 | OBJE | CTIVES | 27 |
| <ol> <li>3.</li> </ol> | | DY DESIGN | |
| ٥. | 3.1. Endpoints | | |
| | 3.1. | Study Design | |
| | 3.3. | Study Treatment | |
| | 3.4. | Duration of Treatment | |
| | 3.5. | Discontinuation Criteria | |
| | 3.6. | Source Data | |
| 4. | SUBJECT POPULATION | | |
| | 4.1. | Number of Subjects and Subject Selection | 30 |
| | 4.2. | Inclusion Criteria | |
| | 4.3. | Exclusion Criteria. | 32 |
| 5. | INVE | STIGATIONAL MEDICINAL PRODUCTS | 34 |
| | 5.1. Randomization and Treatment Codes | | |
| | 5.2. | Description and Handling of Sofosbuvir/Ledipasvir Fixed-Dose Combination | 34 |
| | | 5.2.1. Formulation | |
| | | 5.2.2. Packaging and Labeling | 34 |
| | | 5.2.3. Storage and Handling | |
| | 5.3. | Dosage and Administration of Sofosbuvir/Ledipasvir FDC | |
| | 5.4. | Prior and Concomitant Medications | |
| | 5.5. | Accountability for SOF/LDV FDC | |
| | | 5.5.1. Investigational Medicinal Product Return or Disposal | |
| 6. | STUE | DY PROCEDURES | 38 |
| | 6.1. | Subject Enrollment and Treatment Assignment | |
| | 6.2. | Pretreatment Assessments | |
| | | 6.2.1. Screening Visit (Day -28 to Day -1) | 38 |

| | 6.3. | Randomization | 40 |
|---|---|---|---|
| | 6.4. | Treatment Assessments | 40 |
| | | 6.4.1. Baseline/Day 1 Visit | 40 |
| | | 6.4.2. Week 1 (± 3 days) | 41 |
| | | 6.4.3. Week 2 (± 3 days) | |
| | | 6.4.4. Week 4 (± 3 days) | |
| | | 6.4.5. Week 6 (± 3 days) | |
| | | 6.4.6. Week 8 (± 3 days) | |
| | | 6.4.7. Week 10 (± 3 days) | |
| | | 6.4.8. Week 12 (± 3 days) | |
| | | 6.4.9. Early Termination (ET)/Unscheduled Visit | |
| | 6.5. | Post-Treatment Assessments. | |
| | 0.5. | 6.5.1. Post Treatment Week 4 (± 5 days) | |
| | 6.6. | | |
| | 0.0. | Procedures and Specifications | |
| | | 6.6.2. Medical History | |
| | | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | |
| | | T T | |
| | | - C | |
| | | 6.6.11. Pharmacogenomic (PG) Substudy | |
| | 6.7. | 6.6.13. Health Related Quality of Life Survey | |
| | | • | |
| 7. | ADV | ERSE EVENTS AND TOXICITY MANAGEMENT | 52 |
| | 7.1. | Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events | 52 |
| | | 7.1.1. Adverse Events | 52 |
| | | 7.1.2. Serious Adverse Events | 52 |
| | 7.2. | Assessment of Adverse Events and Serious Adverse Events | 53 |
| | | 7.2.1. Assessment of Causality for Study Drugs and Procedures | 53 |
| | 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Seriou | | |
| | | Adverse Events to Gilead or CRO | |
| | 7.4. | Gilead Reporting Requirements | 55 |
| | 7.5. | Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or | |
| | | Serious Adverse Events | 56 |
| | 7.6. | Subject Stopping Rules | 56 |
| | 7.7. | Special Situations Reports. | 57 |
| | | 7.7.1. Definitions of Special Situations | 57 |
| | | 7.7.2. Instructions for Reporting Special Situations | 57 |
| 8. | STAT | TISTICAL CONSIDERATIONS | 59 |
| | 8.1. | Analysis Objectives and Endpoints | 59 |
| | J | 8.1.1. Analysis Objectives | |
| | | 8.1.2. Primary Endpoint | |
| | | 8.1.3. Secondary Endpoint | |
| | | 8.1.4. Other Endpoints of Interest | |
| | 8.2. | Analysis Conventions. | |
| | | <i>y</i> | |

| | | 8.2.1. | Analysis Sets | 60 |
|---|---|---|---|---|
| | 8.3. | Data H | andling Conventions | 61 |
| | | 8.3.1. | Interim Analysis | 62 |
| | 8.4. | | raphic Data and Baseline Characteristics | |
| | 8.5. Efficacy Analysis | | | |
| | | 8.5.1. | Primary Analysis | |
| | | 8.5.2. | Secondary Analysis | |
| | 8.6. | • | Analysis | |
| | | 8.6.1. | Extent of Exposure | |
| | | 8.6.2. | Adverse Events | |
| | | 8.6.3. | Laboratory Evaluations | |
| | 8.7. | | cokinetic Analysis | |
| | 8.8. Sample Size | | Size | 65 |
| 9. | RESP | ONSIBIL | JTIES | 67 |
| | 9.1. | Investig | gator Responsibilities | 67 |
| | | 9.1.1. | Good Clinical Practice | 67 |
| | | 9.1.2. | Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | |
| | | | Review and Approval | 67 |
| | | 9.1.3. | Informed Consent | |
| | | 9.1.4. | Confidentiality | 68 |
| | | 9.1.5. | Study Files and Retention of Records | 68 |
| | | 9.1.6. | Case Report Forms | |
| | | 9.1.7. | Investigational Medicinal Product Accountability and Return | 70 |
| | | 9.1.8. | Inspections | 70 |
| | | 9.1.9. | Protocol Compliance | 70 |
| | 9.2. | Sponso | r Responsibilities | 71 |
| | | 9.2.1. | Protocol Modifications | 71 |
| | | 9.2.2. | Study Report and Publications | |
| | 9.3. | | vestigator/Sponsor Responsibilities | |
| | | 9.3.1. | Access to Information for Monitoring | |
| | | 9.3.2. | Access to Information for Auditing or Inspections | |
| | | 9.3.3. | Study Discontinuation | |
| 10. | REFE | ERENCES | | 73 |
| 11. | APPE | ENDICES | | 79 |
| | Anno | ndiv 1 | Investigator Signatura Paga | 0.0 |
| | Appendix 1. | | Investigator Signature Page Study Procedures Table | |
| | Appendix 2. | | GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities | |
| | Appendix 3. Appendix 4. | | Pregnancy Precautions, Definition for Female of Childbearing Potential, and | 63 |
| | Appe | nuix 4. | Contraceptive Requirements | 108 |
| | Anne | ndix 5. | Calculation of Historical Control SVR12 for Treatment-naïve Korean Subjects and | 100 |
| | Аррсі | nuix 3. | for Treatment-naïve Chinese Subjects with Chronic GT-1 HCV Infection | 110 |
| | LICTE OF INTERVENTED A DIFFE | | | |
| | | | LIST OF IN-TEXT TABLES | |
| | Table | 1-1. | GS-US-334-0111 Geometric Least-Squares Mean Ratios (90% Confidence | |
| | | | Intervals) for Sofosbuvir, GS-566500, GS-331007, and Ledipasvir Primary PK | |
| | | | Parameters in Japanese versus Caucasian Subjects | |
| | | | GS-US-337-0113 Number (and Percentage) of Subjects with SVR12 | |
| | Table | 5-1. | Disallowed and Concomitant Medications to be used with Caution | 36 |

#### PROTOCOL SYNOPSIS

Gilead Sciences, Inc. 333 Lakeside Drive Foster City, CA 94404, USA

## **Study Title:**

A Phase 3b, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination in Treatment-Naïve and Treatment-Experienced Subjects with Chronic Genotype 1 HCV Infection

IND Number: EudraCT Number: Not applicable Not applicable

NCT02021656

Clinical Trials.gov Identifier:

-----

**Study Centers Planned:** 

Approximately 20 sites in China Approximately 14 sites in Korea Approximately 10 sites in Taiwan

#### **Objectives:**

The primary objectives of this study are:

- To determine the antiviral efficacy of treatment with sofosbuvir (SOF)/ledipasvir (LDV) fixed-dose combination (FDC) as measured by the proportion of subjects with sustained virologic response (SVR) 12 weeks after discontinuation of therapy (SVR12, defined as HCV RNA < lower limit of quantification [LLOQ] 12 weeks post treatment)
- To evaluate the safety and tolerability of SOF/LDV FDC as assessed by review of the accumulated safety data

The secondary objectives of this study are:

- To determine the proportion of subjects who attain SVR at 4 and 24 weeks after discontinuation of therapy (SVR4 and SVR24)
- To evaluate the kinetics of circulating HCV RNA during treatment and after treatment discontinuation
- To evaluate the emergence of viral resistance to SOF and LDV during treatment and after treatment discontinuation

The exploratory objectives of this study are:



## **Study Design:**

International (China, Korea and Taiwan), multicenter, open-label study in treatment-naïve and treatment-experienced adults with chronic genotype 1 HCV infection.

Approximately 180 treatment-naïve and 180 treatment-experienced subjects will receive treatment with SOF 400 mg/LDV 90 mg fixed dose combination (FDC) tablet for 12 weeks.

It is estimated that approximately 200 subjects will be enrolled in China, 80 subjects will be enrolled in Korea, and 80 subjects in Taiwan. Within each country approximately 50% (i.e., n~100 or 40) of subjects will be treatment-naïve and 50% will be treatment-experienced (i.e., n~100 or 40).

Treatment-naïve is defined as having never received treatment for HCV with any interferon (IFN), ribavirin (RBV), or other approved or experimental HCV-specific direct acting antivirals.

Treatment-experienced is defined as:

a) IFN intolerant

Note: Subjects intolerant of Peg-IFN $\alpha$ +RBV+HCV protease inhibitor regimens are included in this category.

- b) Non-response
- c) Relapse/Breakthrough

Note: For treatment-experienced subjects, prior exposure to HCV NS3/NS4A protease inhibitors is permitted.

Up to 20% of subjects enrolled in the study may have compensated cirrhosis at Screening.

Number of Subjects Planned:

Approximately 360 subjects

Target Population: Treatment-naïve and treatment-experienced, chronic genotype 1 HCV

infected adults

Duration of Treatment:

12 weeks

Diagnosis and Main Eligibility Criteria: Chronic genotype 1, HCV infected, male and non-pregnant/non-lactating female subjects, ages 20 years and older, treatment-naïve or treatment-experienced, of whom approximately 20% may have compensated cirrhosis, may be eligible for the study.

Reference Section 4.2 and 4.3 for detailed Inclusion and Exclusion criteria.

Study Procedures/ Frequency: Screening assessments will be completed within 28 days of the Baseline/Day 1 visit. The screening window can be extended to 42 days for subjects requiring liver biopsy or additional HCV genotyping.

Study visits will occur at Screening, Baseline/Day 1, and on-treatment at the end of Weeks 1, 2, 4, 6, 8, 10, and 12. Following the last dose of study medication, all subjects will complete 4-Week and 12-Week Post-Treatment Visits. Subjects with HCV RNA < LLOQ at the 12-Week Post-Treatment Visit will also complete a 24-Week Post-Treatment Visit unless confirmed viral relapse occurs.

Administration of interferon or any HCV-directed treatment, other than the study drug, is prohibited from 12 weeks prior to Screening until completion of the final post-treatment follow-up visit.

Screening assessments include physical examination, height, weight, vital signs, 12-lead electrocardiogram (ECG), medical history, adverse events (AEs), concomitant medications, safety laboratory tests (hematology, chemistry, coagulation, urinalysis), HCV RNA, serology (HIV, HCV, HBV), hemoglobin A1c (HbA1c), assessment of the presence or absence of cirrhosis, liver imaging for HCC (cirrhotics only), serum  $\beta$ -hCG (females of child bearing potential only), thyroid stimulating hormone (TSH), HCV genotyping, IL28B genotyping.

On-treatment assessments include adverse events (AEs), concomitant medications, review of study drug adherence, physical examinations, vital signs, safety laboratory tests, HCV RNA, pharmacokinetic samples, and urine pregnancy tests (females of child bearing potential only).

Single 12-lead ECGs will be collected at Screening, Baseline/Day 1 (prior to study drug administration) and on-treatment visits at the end of Weeks 1 and Week 12.

Weight will be measured at Screening, Baseline/Day 1, on-treatment visit at the end of Week 12, and post-treatment Weeks 12 and 24 visits (as applicable).

Health Related Quality of Life (HRQoL) Survey will be conducted at Baseline/Day 1, on-treatment visits at the end of Weeks 2, 4, 8, and 12, and Post-Treatment Week 4 and 12 visits.

Pregnancy prevention counseling will be addressed with the subject at Baseline/Day 1, on-treatment visit at the end of Week 12, and post-treatment Week 4 visits.

Post-treatment assessments include AEs, concomitant medications, vital signs, safety laboratory tests, HCV RNA, and urine pregnancy tests (females of child bearing potential only).

Samples for viral RNA sequencing/phenotyping will be collected at Baseline/Day 1 and every visit thereafter. Single PK samples will be collected during on-treatment visits for PK analysis of study drug.

Two archive plasma samples will be collected, one at Baseline/Day 1 and the second at the end of treatment visit for potential future biomarker testing. Subjects will have the opportunity to opt out of the archive sample collection. For subjects who provide their additional and specific consent, a blood sample will be collected at the Baseline/Day 1 visit for human pharmacogenomic testing (this sample may be drawn after Baseline/Day 1, if necessary).

Optional Substudies:



| | PPD |
|---|---|
| Test Product, Dose,<br>and Mode of<br>Administration: | SOF/LDV is manufactured as a FDC tablet, consisting of 400 mg SOF and 90 mg LDV, for oral administration. Subjects will take 1 tablet daily with or without food. |
| Reference Therapy, None. Dose, and Mode of Administration: | |
| Criteria for<br>Evaluation: | |
| Safety: | AEs and safety laboratory tests will be collected throughout the study (through the 4-Week Post-Treatment Visit). |
| Efficacy: | Efficacy will be evaluated using scheduled assessments of HCV RNA performed using COBAS® TaqMan® HCV Test, v2.0 for use with the High Pure System or COBAS® AmpliPrep / COBAS® TaqMan® HCV Test, v2.0. |
| Pharmacokinetics: | In China, Korea and Taiwan, a single PK blood sample will be collected at each on-treatment visit for all subjects. PPD If conducted, a target of ~10-15 subjects may be enrolled from each country. Serial PK samples would be collected over 24 hours post-dose. The PK of SOF (and its metabolites GS-566500 and GS-331007) and LDV will be assessed. |
| Statistical Methods: | The primary efficacy endpoint is SVR12 in all enrolled and treated subjects with chronic genotype-1 HCV infection. The primary endpoint will be performed on the Full Analysis Set (FAS). |
| | Treatment-Naïve Subjects |
| | The primary endpoint will be assessed by comparison of the observed SVR12 rate for treatment-naïve subjects with HCV GT-1 infection from Korea and China versus the historical SVR null rate of 49% and 57% respectively (as calculated in Appendix 5) using a two-sided exact one-sample binomial test. |
| | the political trial and the Property Appears appears of the party than the party of |

Taiwan, and overall (i.e., China plus Korea plus Taiwan),

In addition, for each region (i.e., China, Korea or Taiwan), Korea plus

a point-estimate with two-sided 95% exact confidence interval using

A sample size of 40 Korean subjects in the treatment-naïve group will provide at least 90% power to detect a 27% improvement in SVR12 rate from the adjusted historical control rate of 49% using 2-sided exact one-sample binomial test at significant level of 0.05.

A sample size of 100 Chinese subjects in the treatment-naïve group will provide at least 90% power to detect a 17% improvement in SVR12 rate from the historical control rate of 57% using 2-sided exact one-sample binomial test at significant level of 0.05.

In addition, with 40 subjects in Korea (or Taiwan), the 2 sided 95% exact confidence interval for the SVR12 rate will extend at most 32% in length. With 80 subjects (Korea plus Taiwan) in the treatment-naïve group, a two-sided 95% exact confidence interval for the SVR12 rate will extend at most 23% in length. With 100 subjects in China, the 2 sided 95% exact confidence interval for the SVR12 rate will extend at most 20% in length.

## **Treatment-Experienced Subjects**

There is no treatment option available in China, Korea or Taiwan for treatment-experienced patients with GT-1 infection. In the absence of effective antiviral therapy, spontaneous clearance of the HCV is rare. Consequently a nominal SVR rate of 5% is assumed for treatment-experienced subjects.

No statistical hypothesis testing will be performed in treatment-experienced subjects. For each region (i.e., China, Korea or Taiwan), Korea plus Taiwan, and overall (i.e., China plus Korea plus Taiwan), a point-estimate with two-sided 95% exact confidence interval using the binomial distribution (Clopper-Pearson method) will be constructed for the SVR12 rate.

With 40 subjects in Korea (or Taiwan), the 2 sided 95% exact confidence interval for the SVR 12 rate will extend at most 32% in length. With 80 subjects (Korea plus Taiwan) in the treatment-experienced group, a two-sided 95% exact confidence interval for the SVR12 rate will extend at most 23% in length. With 100 subjects in China, the 2 sided 95% exact confidence interval for the SVR12 rate will extend at most 20% in length.

Secondary efficacy endpoints include the proportion of subjects with SVR4, SVR24, breakthrough and relapse; and HCV RNA change from baseline.

All continuous endpoints (except safety endpoints) will be summarized using an 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) by treatment-naïve and treatment-experienced subjects for each region and overall. All categorical endpoints will be summarized by number and percentage of subjects who meet the endpoint definition.

Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data.

This study will be conducted in accordance with the guidelines of Good Clinical Practices (GCPs) including archiving of essential documents.

## GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

° C degrees Celsius
° F degrees Fahrenheit

β-hCG β-human chorionic gonadotropin

AE adverse event

ALT alanine aminotransferase (also SGPT)

ANC absolute neutrophil count

APTT Activated partial thromboplastin time
AST Aspartate aminotransferase (also SGOT)

AUC area under the curve

AUC<sub>tau</sub> area under the plasma concentration versus time curve over the dosing interval

(tau)

BID twice a day

BLQ below the lower limit of quantification

BMI body mass index
BT breakthrough
BW body weight

CFR Code of Federal Regulations

CL<sub>cr</sub> creatinine clearance

 $C_{max} \hspace{1.5cm} \hbox{the maximum observed serum/plasma/peripheral blood mononuclear (PBMC)} \\$ 

concentration of drug

C<sub>tau</sub> Observed drug concentration at the end of the dosing interval (tau)

CRF case report form(s)

CRO Contract (or clinical) research organization

DAA Direct acting antiviral

DCV Daclatasvir dL Deciliter

DNA deoxyribonucleic acid

DSPH Drug Safety and Public Health

ECG Electrocardiogram

ECIRB/IEC Ethics Committee Institutional Review Board/ Independent Ethics Committee

eCRF Electronic case report form(s)

E<sub>max</sub> Maximal effect

ESA Erythropoiesis stimulating agent

eSAE electronic Serious Adverse Event (system)

ESLD End Stage Liver Disease

ET early termination
EU European Union
FAS full analysis set

FDA (United States) Food and Drug Administration

## GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS (CONTINUED)

FDC Fixed Dose Combination

FEV<sub>1</sub> forced expiratory volume in one second GCP Good Clinical Practice (Guidelines)
GCSF Granulocyte colony stimulating factor

GGT gamma glutamyl transferase

GMRs geometric-least squares means ratios

GSI Gilead Sciences, Inc.

GT Genotype (viral)

Hb Hemoglobin

HbA<sub>1c</sub> Hemoglobin  $A_{1c}$ 

HBsAg Hepatitis B virus surface antigen

HBV Hepatitis B virus

HCC Hepatocellular Carcinoma

HCV Hepatitis C virus

HCV Ab Hepatitis C virus antibody
HDPE high-density polyethylene

HIV Human Immunodeficiency Virus

HLGT High-Level Group Term

HLT High-Level Term

HRQoL Health Related Quality of Life (Survey)
ICH International Conference on Harmonisation

IEC Independent Ethics Committee

IFN interferon
IL28B IL28B gene

IMP Investigational Medicinal Product
IND Investigational New Drug (Application)

INR International Normalized Ratio
IRB Institutional Review Board

IUInternational UnitsIUDIntrauterine Device

IV Intravenous

IVDA Intravenous drug abuse

IWRS Interactive Web Response System

kg Kilogram
L Liter
LDV Ledipasvir

LLN lower limit of the normal range LLOQ Lower limit of quantification

## GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS (CONTINUED)

LLT Lower-Level Term LTFU Lost to follow up

Medical Dictionary for Regulatory Activities

Mg Milligram mL Milliliter

mmHg millimeters mercury
NS (3/4A/5A/5B) Non-structural Protein

PBMC peripheral blood mononuclear cell(s)

 Peg-IFNα
 pegylated interferon

 PG
 Pharmacogenomic

 P-gp
 P-glycoprotein

 PI
 Protease inhibitor

 PK
 Pharmacokinetic

 PT
 Preferred Term

 QA
 Quality Assurance

QD once daily (use only in tables)

QTcF QT interval corrected using Fridericia' formula

RBC Red blood cell count

RBV Ribavirin

RNA ribonucleic acid

RVR rapid virologic response
SAE serious adverse event
SD Standard deviation
SF-36 Short-Form-36

SOC Standard of Care or System Organ Class

SOF Sofosbuvir

SOP Standard operating procedure

SUSAR Suspected Unexpected Serious Adverse Reaction

SVR Sustained Virologic Response
TE Treatment-Experienced

TN Treatment-Naïve

TGV Tegobuvir

TND Target not detected TPO thrombopoietin

TSH Thyroid stimulating hormone

 $t^{1/2}$  An estimate of the terinal elimination half-life of the drug in

serum/plasma/PBMC, calculated by dividing the natural log of 2 by the terminal

elimination rate contstant ( $\lambda z$ )

ULN upper limit of the normal range

# GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS (CONTINUED)

US United States

WBC white blood cell count

## 1. INTRODUCTION

## 1.1. Background

#### 1.1.1. HCV Infection

Infection with the hepatitis C virus (HCV) is a serious, progressive, and often life-threatening disease affecting approximately 180 million adults worldwide {21360}. The infection, if untreated, can result in progressive liver fibrosis, cirrhosis, hepatocellular carcinoma (HCC) and end stage liver disease (ESLD). Transmission of HCV infection is parenteral with the majority of infections occurring through administration of contaminated blood products, unsafe medical procedures, intravenous drug use or sexual transmission {8076}. The hepatitis C virus is classified into six major genotypes (GT), i.e., 1-6, with further division to a subtype level (e.g., a, b, c) {21479}. Virologic response rates to currently available therapies vary according to host IL28B genotype, baseline levels of HCV RNA and HCV genotype. The distribution of HCV genotypes and subtypes varies according to geographic region with the most common HCV genotypes in the United States and Europe being GT-1, GT-2 and GT-3. In China GT-1, GT-2 and GT-6 are generally the most common although regional differences in genotype distribution, such as GT-3 in the South, are apparent {24217}. In Korea and Taiwan it is estimated that approximately 50% of infections are associated GT-1b and 50% with GT-2a {24218}, {29246}, {24215}. Genotypes 4, 5 and 6 are most prevalent in the Middle East, South Africa and Southeast Asia respectively {22110}.

Following acute infection approximately 15-20% of patients are able to clear the virus without intervention, however around 80% of patients go on to establish chronic hepatitis C {8076}. Treatment of chronic infection is currently based upon weekly subcutaneous administration of pegylated interferon (Peg-IFNα) with orally administered ribavirin (RBV) for 24 to 48 weeks dependent upon genotype and virologic response. In Caucasians, this treatment regimen affords sustained virologic response rates (SVR) on the order of 42-46% in treatment-naïve patients with GT-1 and 76-82% in patients with GT-2/3 infection {23342}, {23351}. Observed SVR rates using the same interferon (IFN)-based treatment regimens are generally higher in Asian patients. This observation has been largely attributed to a higher proportion of Asian patients (>85%) possessing the host IL28B-CC genotype which confers a favorable virologic outcome following treatment with IFN-containing regimens {22075}, {24243}, {22156}, {21337}, {22098}. Although relatively high SVR rates can be achieved in Asian patients with IFNα+RBV, the safety and tolerability of IFN-containing regimens is sub-optimal. Contraindications to IFN preclude its use by a significant number of patients {22156} while management of adverse effects commonly results in dose reductions and may lead to treatment discontinuation. Safety and tolerability are particularly problematic in an aging population with chronic hepatitis C. Moreover, lower SVR rates are also observed in older patients {24406}.

Recently, first generation protease inhibitors (PI) (i.e., telaprevir (TVR) and boceprevir (BCV)) have been approved in certain countries for use in patients with GT-1 infection when combined with Peg-IFN $\alpha$ +RBV. The Peg-IFN $\alpha$ +RBV+PI regimens have incrementally improved SVR rates in GT-1 treatment-naïve patients to approximately 70%; however, they are associated with

significant safety and tolerability concerns  $\{17996\}$ ,  $\{17492\}$ . Moreover, Peg-IFN $\alpha$ +RBV+PI regimens are not currently available in Korea, Taiwan or China and, consequently, patients with GT-1 infection who fail to respond to Peg-IFN $\alpha$ +RBV have no current treatment options.

#### 1.1.2. HCV Infection in Korea

In Korea, chronic HCV infection is one of the leading causes of chronic liver disease and hepatocellular carcinoma (HCC) {24211}. The age-standardized prevalence of HCV antibody (HCV Ab) in patients greater than 40 years of age is reported to be on the order of 1.3% which equates to around 193,000 people {24215}. The prevalence of HCV infection increases with age and peaks in those individuals aged 60 years and older {24211}. The majority of infections occurred via contaminated blood transfusions prior to the introduction of blood-donor HCV Ab screening in 1991 {24216}. Consequently the majority of patients with chronic hepatitis C in Korea are elderly {24215} and are more likely to have progressive liver disease. HCV infection is more closely associated with HCC in the elderly Korean patients than are HBV infection and alcoholism {24210}, {24208}. Since the decline of transfusion-related hepatitis C the majority of new infections are behavior-related. Of particular note is the practice of acupuncture for chronic illnesses including joint disease, pain, sequelae of trauma and other conditions non-responsive to conventional therapies. Shin et al reported results of a case study in which 34.1% of men and 62.9% of women in rural Korea reported multiple acupuncture procedures with the associated risk fraction for HCV infection being 38% for men and 55% for women {24214}. Intravenous drug abuse (IVDA) is not thought to be a major contributor to the overall prevalence of HCV infection in Korea however this route of infection may contribute in young adults and those living in harbor cities on the southern and western coasts {24209}, {24211}. The predominant HCV genotypes in Korea are GT-1b and GT-2a which are roughly present in equal proportions and combined account for around 80-90% of infections {24216}, {24215}, {24209}. Host IL28B genotype has been widely reported as a predictor of virologic response to interferon (IFN)-based therapies for chronic HCV infection {22075}. The IL28B-CC genotype which confers a favorable virologic outcome to IFN-based therapy predominates in Korea with approximately 80-90% of patients with this genotype {24212}, {24238}. Consequently the sustained virologic response rates in Korean clinical trials evaluating Peg-IFNα+RBV in treatment-naïve GT-1 infection are on the order of 55-70% following 48 weeks of therapy {24211}, {24595}, {24387}, {24385}, {24237}, {24404}, {24388}. Although relatively high rates of virologic response are achievable with Peg-IFNα+RBV in treatment-naïve Korean patients due to the high proportion of IL28B CC genotype, Heo et al {24236} recently reported a significant difference in SVR rate observed in a clinical trial cohort versus that observed in clinical practice based upon 'Intention To Treat' (ITT) analysis; 81% (21/26) versus 55% (58/106). Although no difference was observed in the SVR rates between the clinical trial cohort and the clinical practice cohort according to per protocol analysis, the ITT is important since it more likely reflects the observed SVR in clinical practice across the country. The authors attribute the lower ITT SVR rate in the clinical practice cohort to decreased adherence to assigned therapy including dose reduction for clinical and laboratory adverse events. As previously described, the highest prevalence rates for HCV Ab in Korean patients are in those individuals aged 60 years and older. These elderly patients are more likely to be treatment-experienced and have progressive liver disease. Comorbid conditions (e.g., diabetes and cardiovascular disease) are common in this population and pose significant

challenges to the use of Peg-IFN $\alpha$ +RBV therapy. As this group of patients continues to age the proportion of patients with chronic hepatitis C who will develop complications, including liver cirrhosis, HCC and ESLD is significant; {22077}. In addition, it is important to consider the proportion of patients who are ineligible for, intolerant of, or unwilling to receive Peg-IFN $\alpha$ +RBV who have no currently available antiviral treatment options {21256}. This also applies to patients who have previously failed to respond to Peg-IFN $\alpha$ +RBV therapy. Although Peg-IFN $\alpha$ +RBV can achieve high rates of SVR in treatment-naïve patients with chronic HCV infection when assigned therapy is tolerated, there is an unmet medical need for effective, safe, well-tolerated, all oral therapies that can be used in an aging patient population in Korea.

#### 1.1.3. HCV Infection in Taiwan

Taiwan has one of the highest prevalence rates of chronic hepatitis C in North-East Asia. In a nationwide survey conducted between 1996 and 2005 involving over 164,000 participants in out-reach community-based hepatitis screening programs the HCV seroprevalence was estimated to be 4.4% {24235}. The study reported an approximately equal seroprevalence in males (4.5%) and females (4.3%). Importantly seroprevalence varied geographically with certain areas of hyperendemicity such as Miaoli and Chiavi Counties where the age-adjusted seroprevalence was reported to be 7.6% and 6.1% respectively. The proportion of subjects with HCV antibodies progressively increased after the age of 20 years. The predominant routes of transmission are thought to be iatrogenic in nature including history of blood transfusion, medical injections and acupuncture {29245}, {29248}. Historically, glucose supplements, vitamins, and treatments for minor medical conditions have often been administered by injection. Prior to 1980 reusable syringes were commonly used particularly in rural areas with poor sterilization techniques likely contributing to the spread of HCV infection. After 1980, the rate of HCV infection was likely reduced following the introduction of disposable syringes. This may in part explain the higher prevalence of HCV infection in the elderly population in Taiwan. It has also been postulated that inhabitants of communities with high rates of HCV infection may have been repeatedly exposed to a common reservoir of infection contributing to the establishment of hyperendemic areas {29245}.

As previously described for Korea, the predominant HCV genotypes in Taiwan are GT-1b and GT-2a which are present in similar proportions and account for around 80-90% of all infections  $\{29247\}$ ,  $\{24218\}$ ,  $\{29246\}$ . The IL28B-CC host genotype conferring favorable virologic outcome to IFN-based therapy predominates with approximately 80-90% of patients with this genotype  $\{22075\}$ ,  $\{24241\}$ . As a consequence the SVR rates in Taiwanese clinical trials evaluating Peg-IFN $\alpha$ +RBV in GT-1 infection are approximately 49-56% and 76-80% in treatment-naïve patients receiving 24 weeks and 48 weeks of treatment respectively  $\{24410\}$ ,  $\{24382\}$ . However, as previously described in Taiwan the seroprevalence of HCV antibodies increases with age with the highest rates observed in those 60 years and older  $\{24235\}$ . The use of currently available therapy is problematic in the elderly due to contraindications to IFN and RBV and comorbidities such as cardiovascular disease and diabetes. In Taiwan for treatment-naïve patients with GT-1 infection aged  $\geq$ 65 years the SVR rate for Peg-IFN $\alpha$ +RBV administered for 48 weeks has been reported to be 51.9%  $\{24390\}$ . The elderly patient population is more likely to have progressive liver disease and be at higher risk for the development of HCC and ESLD. For GT-1 infection

the SVR rates for Taiwanese age-matched patients with HCC (post-curative management) and cirrhosis are reported to be 33% and 55% respectively {24240}. The safety, tolerability and efficacy of IFN+RBV therapy is suboptimal in this population. Finally, there are no currently available treatment options for those patients who are ineligible for, intolerant of, or who have previously failed to respond to IFN+RBV therapy.

#### 1.1.4. HCV Infection in China

Reports indicate that around 2% of the population in China, or approximately 27 million people, may be infected with the hepatitis C virus {19682},{24217},{25129}. Approximately 68% of patients are infected with HCV GT-1b, 14% with GT-2, 4% with GT-3 and 13% with GT-6 {19682},{24217}. GT-1 and GT-2 infection are generally more common in older patients whereas GT-3 and GT-6 are more frequent in younger adults. This observation may be related to the mode of HCV transmission, with GT-1/GT-2 commonly acquired through prior blood transfusion and GT-3/GT-6 associated with IVDA {25094}.

Risk factors for HCV infection are similar to those reported in other parts of the world {25095}. Of note, however, is the reported risk of acquiring transfusion-related HCV infection which is on the order of 1 in 40,000-60,000 donations {25093}. Such high rates of transfusion-related hepatitis C have been attributed in part to the practice of paid blood donation. Following introduction of mandatory HCV screening of blood/blood products in the 1990's and the implementation of the blood donation law in 1998, the incidence of post-transfusion hepatitis C has been significantly reduced {24392, 25127}. The association of GT-1 infection with blood transfusion and the timing of the new requirements related to blood donation may in part explain the higher GT-1 infection rates in the elderly. Since the introduction of blood-bank screening, the predominant mode of new HCV infection is now intravenous drug use (IDU).

The recommended treatment regimen for treatment-naïve patients with HCV GT-1 in China according to the Chinese Society of Hepatology  $\{24428\}$  is subcutaneous or intramuscular administration of IFN $\alpha$  or Peg-IFN $\alpha$  plus orally administered RBV for 24 to 48 weeks according to baseline viral load and virologic response. These recommendations are aligned with those by the APASL Consensus Committee  $\{24699\}, \{22156\}$ . SVR rates in China for GT-1have been reported to be on the order of 44% to 70%  $\{24797\}, \{13261\}, \{24391\}$ .

A significant number of patients in China are in the  $3^{rd}$ - $4^{th}$  decade of infection and have progressive liver disease. The use of IFN $\alpha$ +RBV therapy in the elderly is problematic. Comorbid conditions are common (eg, cardiovascular disease, diabetes, mental anomaly, decreased renal function) and may preclude IFN $\alpha$  use {24428} {22156} {24398}. Older patients generally report a higher frequency of adverse events and of greater severity compared to younger patients. Lower levels of treatment adherence are also observed. These factors contribute to overall lower SVR rates observed with IFN-based therapy in the elderly {24390}. As patients continue to age, the number developing hepatic complications including cirrhosis, HCC and ESLD will be significant {22077}.

The use of IFN $\alpha$ -based therapy is also problematic in the IVDA population. The risk for developing severe IFN $\alpha$ -related psychiatric events including depression, suicidal ideation,

cognitive disturbances, psychotic symptoms, fatigue and habit relapse is high. Adherence to therapy may be low and effective treatment requires multidisciplinary support {25091}.

A significant number of patients are ineligible for, or unwilling to undergo treatment with IFN-based therapy. For these patients, there are presently no available therapeutic options available

## **1.1.5. Summary**

There is a need for early intervention and eradication of HCV infection to reduce the burden of progressive liver disease including of HCC and ESLD. While early introduction of effective antiviral therapy is critical in order to reduce the potential future burden of advanced liver disease, safe and effective antiviral therapies that can be used in elderly patients with advanced disease is of paramount importance today. Gilead Sciences is developing the all-oral, interferon- and ribavirin-free SOF/LDV FDC regimen to address this need in Chinese, Korean and Taiwanese patients with chronic genotype-1 HCV infection.

# 1.2. Sofosbuvir (formerly GS-7977) and Ledipasvir (formerly, GS-5885) Fixed Dose Combination

Sofosbuvir/Ledipasvir fixed dose combination (FDC) combines two HCV specific DAA agents into a single tablet for the treatment of chronic HCV infection. More than 2500 subjects have received treatment with this combination tablet to date.

Sofosbuvir (SOF), formerly GS-7977, is a nucleotide analog that is a potent and selective inhibitor of NS5B-directed HCV replication. Over 4,000 subjects have received SOF containing regimens to date, from single doses up to repeat dosing for 24 weeks.

Ledipasvir (LDV), formerly GS-5885, is a novel HCV NS5A inhibitor that has demonstrated potent anti-HCV activity against genotype (1a and 1b) HCV infection. More than 1000 HCV infected subjects have been dosed with LDV in Phase 2 clinical studies, and over 700 subjects have been dosed with LDV for over 12 weeks.

#### 1.2.1. General Information

For further information on SOF/LDV FDC and the individual components, refer to the Investigator's Brochure (IB) for sofosbuvir/ledipasvir fixed-dose combination including:

- In Vitro Anti-HCV Activity
- Nonclinical Pharmacokinetics and In Vitro Metabolism
- Nonclinical Pharmacology and Toxicology
- Clinical Experience

## 1.2.2. Summary of Additional Clinical Experience with Sofosbuvir and Ledipasvir

## 1.2.2.1. GS-US-334-0111 Pharmacokinetic Bridging Study in Japanese Subjects

To support the conduct of clinical studies in Japan, a PK bridging study was conducted in accordance with ICHE5 to compare the safety, tolerability and PK profile in Japanese and Caucasian subjects following single-dose administration of SOF at the 200 mg, 400 mg (the intended therapeutic dose) and 800 mg dose levels. This study also evaluated the pharmacokinetic parameters of the 400 mg dose of SOF and the 90 mg dose of LDV administered as a single dose of the SOF/LDV FDC. This study was conducted in the United States.

The study enrolled Japanese and Caucasian subjects with an approximately even distribution of healthy males and healthy, non-pregnant, non-lactating females between 18–45 years, inclusive, with a body mass index (BMI)  $18 \le BMI \le 30$ . Japanese subjects must have been born in Japan, not lived outside Japan for more than 10 years, could trace maternal and paternal Japanese ancestry of parents and grandparents, and their lifestyle, including diet, had not significantly changed since leaving Japan. Caucasian subjects must not have been of Japanese or Asian descent; those with parents or grandparents born in Japan or in any Asian country were excluded.

Eligible subjects received one dose of study treatment on Day 1 corresponding to their assigned group. Each group comprised 8 Japanese and 8 Caucasian subjects and received SOF at either the 200 mg, 400 mg or 800 mg dose levels (Groups 1-3), or 400 mg SOF + 90 mg LDV administered as a single dose of the SOF/LDV FDC (Group 4). Safety was assessed by evaluation of vital signs, 12-lead ECGs, and adverse events. Plasma and urine samples were collected at selected time points to assess the PK of SOF, its metabolites GS-566500 and GS-331007, and LDV.

SOF and SOF/LDV FDC were well tolerated in this study.

Pharmacokinetic (plasma) results are in Table 1-1.

Table 1-1. GS-US-334-0111 Geometric Least-Squares Mean Ratios (90% Confidence Intervals) for Sofosbuvir, GS-566500, GS-331007, and Ledipasvir Primary PK Parameters in Japanese versus Caucasian Subjects

| | SOF 200 mg<br>% GLSM Ratio<br>(90% CI) | SOF 400 mg<br>% GLSM Ratio<br>(90% CI) | SOF 800 mg<br>% GLSM Ratio<br>(90% CI) | SOF/LDV FDC<br>(400 mg/90 mg)<br>% GLSM Ratio<br>(90% CI) |
|---|---|---|---|---|
| SOF PK Parameter | r | | | |
| AUC <sub>last</sub> (ng•h/mL) | 97.02 | 122.62 | 106.20 | 90.52 |
| | (63.62, 147.96) | (92.54, 162.47) | (82.63, 136.49) | (54.44, 150.50) |
| AUC <sub>inf</sub> (ng•h/mL) | 97.30 | 121.98 | 106.27 | 90.77 |
| | (64.77, 146.16) | (92.30, 161.20) | (82.84, 136.33) | (54.90, 150.07) |
| C <sub>max</sub> (ng/mL) | 101.56 | 107.05 | 96.37 | 93.82 |
| | (62.88, 164.02) | (76.31, 150.18) | (62.23, 149.23) | (64.53, 136.42) |
| GS-566500 PK Par | ameter | | | |
| AUC <sub>last</sub> (ng•h/mL) | 158.37 | 149.64 | 125.17 | 114.13 |
| | (119.80, 209.34) | (117.13, 191.17) | (103.74, 151.03) | (78.15, 166.67) |
| AUC <sub>inf</sub> (ng•h/mL) | 153.51 | 147.47 | 124.39 | 113.27 |
| | (117.65, 200.30) | (116.45, 186.74) | (103.30, 149.79) | (78.24, 163.98) |
| C <sub>max</sub> (ng/mL) | 154.48 | 138.62 | 117.59 | 130.16 |
| | (116.12, 205.51) | (108.12, 177.72) | (98.72, 140.06) | (93.88, 180.44) |
| GS-331007 PK Par | ameter | | | |
| AUC <sub>last</sub> (ng•h/mL) | 80.29 | 94.44 | 82.32 | 85.63 |
| | (64.62, 99.77) | (78.30, 113.90) | (71.98, 94.16) | (63.56, 115.36) |
| AUC <sub>inf</sub> (ng•h/mL) | 82.37 | 95.93 | 83.68 | 85.40 |
| | (67.59, 100.36) | (80.14, 114.82) | (74.25, 94.30) | (64.04, 113.89) |
| C <sub>max</sub> (ng/mL) | 72.72 | 113.48 | 102.44 | 94.34 |
| | (57.86, 91.40) | (91.12, 141.32) | (73.52, 142.73) | (68.03, 130.82) |
| LDV PK Parameter | | | | |
| AUC <sub>last</sub> (ng•h/mL) | _ | _ | _ | 106.07<br>(68.95, 163.18) |
| AUC <sub>inf</sub> (ng•h/mL) | _ | _ | _ | 106.66<br>(69.13, 164.59) |
| C <sub>max</sub> (ng/mL) | | _ | _ | 125.63<br>(83.83, 188.26) |

No clinically significant differences in the PK of SOF, its metabolites GS-566500 and GS-331007, or LDV were observed between Japanese and Caucasian subjects. The safety and pharmacokinetic profiles support the use of SOF 400 mg or SOF/LDV FDC (400 mg/90 mg) in Japanese and non-Japanese subjects.

## 1.2.2.2. Phase 3 International Registration Studies with SOF/LDV FDC

The SOF/LDV phase 3 international registration program consists of 3 clinical studies for which data are available: GS-US-337-0102 (ION-1), GS-US-337-0109 (ION-2), and GS-US-337-0108 (ION-3). Studies GS-US-337-0102 and GS-US-337-0109 are evaluating treatment with SOF/LDV±RBV for 12 or 24 weeks in treatment-naive and treatment-experienced subjects, respectively, who are infected with genotype 1 HCV. Both studies enrolled up to 20% of HCV-infected subjects who had documented compensated cirrhosis. ION-3 is evaluating SOF/LDV±RBV treatment for 8 weeks and SOF/LDV treatment for 12 weeks in noncirrhotic treatment-naive subjects with genotype 1 HCV infection.

Across all studies, SOF/LDV demonstrated a high degree of efficacy with point estimates for SVR12 > 93% in subjects with genotype 1 HCV infection. The addition of RBV to the SOF/LDV regimen did not impact the SVR rate.

Across the SOF/LDV Phase 3 studies, treatment with SOF/LDV was generally safe and well tolerated. The 3 most frequently occurring AEs were fatigue, headache, and nausea. A higher incidence of each event was reported in subjects receiving SOF/LDV+RBV compared with subjects receiving SOF/LDV: fatigue (38.0% vs. 22.2%), headache (26.1% vs. 20.6%), and nausea (17.4% vs. 10.4%). The most common Grade 3 or 4 chemistry laboratory abnormalities across all treatment groups were increased lipase (1.7%) and increased serum glucose (1.5%). In subjects with Grade 3 or 4 increased lipase, no case was associated with clinical signs or symptoms of pancreatitis. Among subjects who experienced a Grade 3 or 4 increased serum glucose, all subjects had a history of diabetes, were taking diabetes medication, or had glucose intolerance (denoted by HbA1c > 6.0% at screening).

## 1.2.2.3. Study GS-US-337-0113 SOF/LDV FDC Study in Japan

An open-label, randomized, phase 3b study (GS-US-337-0113) is also being conducted in Japan to assess the efficacy and safety of 12 weeks of SOF/LDV with or without RBV in treatment-naive (TN) and treatment-experienced (TE) subjects with genotype 1 HCV infection.

A total of 341 subjects (166 treatment-naïve and 175 treatment-experienced) were randomized (1:1) to receive treatment. The majority of subjects are female (58%), and all are Japanese. The majority of subjects have genotype 1b HCV infection (97%), non-CC IL28B alleles (52%), high baseline viral load (99% had HCV RNA  $\geq$  5 log<sub>10</sub> IU/mL), 22% had liver cirrhosis at baseline, and 33% were 65 years of age or older.

SVR12 was achieved by 100% (171/171) of subjects receiving SOF/LDV for 12 weeks and by 98% (167/170) subjects receiving SOF/LDV+RBV for 12 weeks (Table 1-2). The study met its primary endpoint of superiority compared to a predefined historical SVR12 rate. Factors that have historically been predictive of or associated with lower rates of SVR (including age ≥65 years, cirrhosis, and prior treatment failure) had no impact on SVR12 rates in this study. Three subjects who received SOF/LDV+RBV did not achieve SVR12: 1 subject relapsed after discontinuation of therapy, 1 patient discontinued therapy after 1 week of treatment due to rash and 1 patient died during the study.

| | Treatment-Naive | | Treatment-Ex | perienced |
|---|---|---|---|---|
| | SOF/LDV<br>12 Weeks<br>(N=83) | SOF/LDV+RBV<br>12 Weeks<br>(N=83) | SOF/LDV<br>12 Weeks<br>(N=88) | SOF/LDV+RBV<br>12 Weeks<br>(N=87) |
| Overall SVR12 | 83/83 (100%) | 80/83 (96%) | 88/88 (100%) | 87/87 (100%) |

Table 1-2. GS-US-337-0113 Number (and Percentage) of Subjects with SVR12

Treatment with SOF/LDV±RBV was generally well tolerated. Most AEs were mild or moderate in severity. The addition of RBV to the SOF/LDV treatment regimen resulted in increased rate of observed AEs (64% of subjects who received SOF/LDV and 75% of those who received SOF/LDV+RBV). The most commonly reported AEs in the RBV-free group were nasopharyngitis, headache, and malaise. The most commonly reported AEs in the SOF/LDV+RBV group were nasopharyngitis, anemia, headache and rash. Nasopharyngitis was thought to be related to the winter season during which the study took place. Two subjects, both in the SOF/LDV+RBV group, permanently discontinued study treatment due to an AE.

Consistent with the expected toxicity profile of RBV, decreases from baseline in hemoglobin and lymphocytes, and increases in reticulocytes and platelets and total bilirubin were observed in the SOF/LDV+RBV 12 Week group.

## 1.3. Rationale for This Study

This Phase 3b study is designed to evaluate the efficacy and safety of the SOF/LDV FDC tablet administered for 12 weeks in treatment-naïve and treatment-experienced subjects with chronic genotype 1 HCV infection. Up to 20% of subjects enrolled in the study may have compensated cirrhosis at screening.

As previously described in Sections 1.1.2 and 1.1.3 in there is a significant unmet medical need in China, Korea and Taiwan for simple, well-tolerated, IFN-free, all-oral antiviral regimens for the treatment of chronic HCV infection. The current standard of care (Peg-IFN $\alpha$ +RBV) for these patients in China, Korea and Taiwan is associated with significant toxicity, with many patients unwilling to be treated with these regimens. There also exists substantial numbers of patients who cannot receive Peg-IFN $\alpha$  due to relative or absolute contraindications {20450}, {17893}, {17893}, {15573}, {17892}, {3291}.

Gilead has developed an FDC consisting of SOF with LDV, 2 well-tolerated, potent, once-daily antiviral agents in late phase clinical development. Based on Phase 2 data, the SOF/LDV FDC has the potential to be a simple and highly effective all-oral, once daily treatment regimen for chronic genotype 1 HCV infection, after 12 weeks of treatment.

In the Phase 3 ION studies, the same SOF/LDV FDC regimen proposed for this study in China, Korea and Taiwan was evaluated in patients with HCV GT-1 infection. SVR12 rates following SOF/LDV for 12 weeks greater than 93% were observed in treatment-naïve subjects with and without cirrhosis (Studies GS-US-337-0102, GS-US-337-0108). In treatment-experienced

subjects in GS-US-337-0109, the SVR12 rate was 94% (n=102/109) overall, with 95% of subjects without cirrhosis achieving SVR12 and 86% of those with cirrhosis achieving SVR12. In Japanese subjects with chronic genotype 1 HCV infection, the SVR12 rate was 100% in both treatment naïve (n=83) and treatment-experienced (n=88) patients following treatment with SOF/LDV for 12 weeks.

Current data for the SOF/LDV FDC indicates the regimen to be safe, well-tolerated and associated with high degrees of antiviral efficacy, supporting the conduct of the proposed Phase 3 study in Chinese, Korean and Taiwanese subjects with GT-1 chronic hepatitis C.

#### 1.4. Rationale for Dose Selection of SOF/LDV FDC

Gilead has developed a fixed-dose combination (FDC) tablet consisting of SOF 400 mg with LDV 90 mg, 2 well-tolerated, potent, once-daily antiviral agents. SOF 400 mg is the marketed dose of SOF in the US and Europe for the treatment of HCV-infection and as such, has been selected for co-formulation with LDV. LDV 90 mg was selected for co-formulation with SOF based on safety, PK and antiviral activity data (studies GS-US-256-0102 and GS-US-248-0120). Study GS-US-256-0102 established the anti-HCV activity of LDV and indicated that the exposures achieved following administration of the 30 mg dose provides >95% of maximal antiviral response in GT 1a HCV infected subjects. It was also observed that 30 mg or greater of LDV likely provided coverage of some drug related mutations that doses less than 30 mg did not, based on an analysis of NS5A mutants that arose in response to exposure to LDV. Therefore, 30 mg and 90 mg of LDV were selected for further clinical evaluation. In Study GS-US-248-0120, 30 mg of LDV was compared to 90 mg of LDV, on a background of 3 other antivirals, vedroprevir (VDV, formerly GS-9451, PI), tegobuvir (formerly GS-9190, NNI), and RBV. Based on a breakthrough rate in the 90 mg arms of 12% compared to a 27% breakthrough rate in the 30 mg arm, 90 mg LDV was selected for further clinical development.

The fixed-dose combination tablet (FDC) of sofosbuvir/ledipasvir 400 mg/90 mg with or without RBV has demonstrated favorable safety and efficacy profiles in over 2500 HCV-infected subjects across different patient populations in Phase 2 and 3 trials. These doses represent the proposed marketed doses of ledipasvir and sofosbuvir that are currently under regulatory review in the US, EU and certain other countries worldwide.

#### 1.5. Overall Risk/Benefit Assessment

The SOF/LDV FDC product combines a potent HCV nucleotide NS5B inhibitor and a potent HCV NS5A inhibitor.

The potential benefits of SOF/LDV FDC for the treatment of chronic HCV are:

- Greater antiviral efficacy (i.e., rapid and durable eradication of HCV) compared to the current standard of care (Peg-IFN $\alpha$  +RBV)
- A reduction in the AEs currently associated with the use of Peg-IFN $\alpha$ +RBV

- A simple, well-tolerated regimen to replace the current complex, response-guided Peg-IFNα +RBV regimens.
- The potential benefit of a shortened SOF/LDV FDC therapy of 12 weeks is a decrease in the burden of treatment for both patients and physicians, through a reduction in the overall number of patient visits.

The safety profile of SOF includes more than 3000 chronic HCV-infected subjects that have been administered over 12 weeks of SOF in combination with a DAA, Peg-IFN $\alpha$ , with or without RBV. No clinical safety issues related to SOF have been identified to date. The safety profile of LDV includes over 1000 chronic HCV-infected subjects, of whom over 700 have been administered more than 12 weeks of LDV, which was given in combination with other DAAs, Peg-IFN $\alpha$ , with or without RBV. No clinical safety issues related to LDV have been identified to date

Furthermore, there is no expectation of significant overlapping or new, unexpected toxicities upon administration of SOF/LDV together as an FDC. To date, the SOF/LDV FDC  $\pm$  RBV has been administered to over 2500 HCV infected subjects in phase 2/3 trials. No clinical safety issues related to the SOF/LDV FDC have been identified to date.

During the conduct of the study the Sponsor will perform ongoing safety data review.

In summary, there is no currently approved all-oral treatment available for HCV-infected patients. This study will support the registration of the SOF/LDV FDC in treatment-naïve and treatment-experienced Chinese, Korean and Taiwanese subjects with chronic genotype 1 HCV infection including those with compensated cirrhosis.

## 1.6. Compliance

This study will be conducted in compliance with this protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements.

## 2. OBJECTIVES

The primary objectives of this study are:

- To determine the antiviral efficacy of treatment with sofosbuvir (SOF)/ledipasvir (LDV) fixed-dose combination (FDC) as measured by the proportion of subjects with sustained virologic response (SVR) 12 weeks after discontinuation of therapy (SVR12, defined as HCV RNA < lower limit of quantitation [LLOQ] 12 weeks post treatment)</li>
- To evaluate the safety and tolerability of SOF/LDV FDC as assessed by review of the accumulated safety data

The secondary objectives of this study are as follows:

- To determine the proportion of subjects who attain SVR at 4 and 24 weeks after discontinuation of therapy (SVR4 and SVR24)
- To evaluate the kinetics of circulating HCV RNA during treatment and after treatment discontinuation
- To evaluate the emergence of viral resistance to SOF and LDV during treatment and after treatment discontinuation

The exploratory objectives of this study are:



## 3. STUDY DESIGN

## 3.1. Endpoints

The primary endpoints of this study are:

- The primary efficacy endpoint is SVR12 (HCV RNA <LLOQ 12 weeks after discontinuation of therapy) in the Full Analysis Set (FAS) population.
- The primary safety endpoint is any AE leading to permanent discontinuation of study drug.

Secondary endpoints of this study include:

• Secondary efficacy endpoints include the proportion of subjects with: HCV RNA < LLOQ at 4 and 24 weeks after discontinuation of therapy (SVR4 and SVR24); viral breakthrough; relapse; and HCV RNA change from baseline.

#### 3.2. Study Design

This will be an international (China, Korea and Taiwan), multicenter, open-label study in treatment-naïve and treatment-experienced adults with chronic genotype 1 HCV infection.

It is estimated that approximately 200 subjects will be enrolled in China, 80 subjects will be enrolled in Korea and 80 subjects in Taiwan for a total of 360 enrolled subjects. Within each country approximately 50% (i.e.,  $n\sim100$  or 40) of subjects will be treatment-naïve and 50% will be treatment-experienced (i.e.,  $n\sim100$  or 40).

Up to 20% of subjects enrolled in the study may have compensated cirrhosis at Screening.

## 3.3. Study Treatment

Approximately 180 treatment-naïve and 180 treatment-experienced subjects will receive treatment with SOF 400 mg/LDV 90 mg fixed dose combination (FDC) tablet for 12 weeks.

#### 3.4. **Duration of Treatment**

All subjects will complete screening, on-treatment, and post-treatment assessments. Screening assessments will be completed within 28 days of the Baseline/Day 1 visit or within 42 days if a liver biopsy or additional HCV genotyping is required. All subjects will receive treatment for 12 weeks. All subjects will complete a 4-week and 12-week Post-Treatment visit. Subjects with HCV RNA < LLOQ at the 12-Week Post-Treatment visit will also complete a 24-Week Post-Treatment visit unless confirmed viral relapse occurs.

The assessments performed at each visit are described in Section 6.

## 3.5. Discontinuation Criteria

When medically feasible, the Medical Monitor must be consulted prior to the premature discontinuation of treatment in a given subject.

Study drug must be discontinued in the following instances:

- Unacceptable toxicity, as defined in Section 7 of the protocol, or toxicity that, in the judgment of the investigator, compromises the ability to continue study-specific procedures or is considered to not be in the subject's best interest
- Pregnancy of female subject

The following on-treatment virologic response-based treatment stopping criteria will be utilized:

- Confirmed HCV RNA ≥ LLOQ after 2 consecutive HCV RNA < LLOQ
- Confirmed > 1 log<sub>10</sub> increase in HCV RNA from nadir
- HCV RNA  $\geq$  LLOQ through 8 weeks of treatment

Confirmation should be performed as soon as possible and must occur no later than 2 weeks after an initial observation indicating virologic failure during the on-treatment phase.

All subjects will complete the 4-Week and 12-Week Post-treatment visits. Subjects with HCV RNA < LLOQ at the 12-week Post-treatment visit will return for the 24-week Post-treatment visit, unless confirmed viral relapse occurs. Study drug may be discontinued in the following instances:

- Significant protocol violation
- Subject request to discontinue for any reason; it is important to determine whether the withdrawal of consent is primarily due to an AE, lack of efficacy, or other reason
- Discontinuation of the study at the request of Gilead, regulatory agency or an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

If a subject meets discontinuation criteria during treatment, an Early Termination (ET) visit will be required (Section 6.4.9). Following completion of the Early Termination visit, all subjects must complete the 4-week and 12-week Post-Treatment visits. All patients with HCV RNA < LLOQ at the 12-week Post-Treatment visit must return to the clinic for 24-week Post Treatment assessments, unless confirmed viral relapse occurs.

#### 3.6. Source Data

A Health Related Quality of Life survey, Short-Form-36 (SF-36) will be completed by subjects at various timepoints during the study and be used as source data. The subject should read the questionnaire by himself/herself and write/mark answers directly onto the questionnaire.

## 4. SUBJECT POPULATION

## 4.1. Number of Subjects and Subject Selection

Approximately 360 subjects will be enrolled in this study with approximately 180 treatment-naïve subjects and approximately 180 treatment-experienced subjects. Up to 20% of subjects enrolled in the study may have compensated cirrhosis at screening.

In order to manage the total study enrollment, Gilead Sciences, Inc., at its sole discretion, may suspend screening and/or enrollment at any site or study-wide at any time.

## 4.2. Inclusion Criteria

Subjects must meet *all* of the following inclusion criteria to be eligible for participation in this study.

- 1) Willing and able to provide written informed consent
- 2) Male or female, age  $\geq$  20 years
- 3) Body weight  $\geq$  40 kg
- 4) HCV RNA  $\geq 10^4$  IU/mL at Screening
- 5) Ability to categorize as treatment-naïve or treatment-experienced, defined below:
  - a) HCV treatment-naïve, as defined as no prior exposure to any IFN, or other approved or experimental HCV-specific direct-acting antiviral agent; OR
  - b) HCV treatment-experienced with medical records that include sufficient detail of prior IFN-based treatment to allow for categorization of prior response as either:
    - *i)* Intolerant: Subject discontinued treatment due to development or significant worsening of an adverse event associated with HCV treatment.
    - ii) Non-Response: Subject did not achieve undetectable HCV RNA levels while on treatment
    - iii) Relapse/Breakthrough: Subject achieved undetectable HCV RNA levels during treatment or within 4 weeks of the end of treatment, but did not achieve a sustained virologic response (SVR)

Treatment-experienced subjects must not have discontinued prior treatment due to non-compliance with treatment.

- 6) Genotype 1 HCV at Screening as determined by the Central Laboratory. Any non-definitive results will exclude the subject from study participation
- 7) Confirmation of chronic HCV infection documented by either:
  - a) A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit, or

- b) A liver biopsy performed prior to the Baseline/Day 1 visit with evidence of chronic HCV infection
- 8) Cirrhosis determination [up to 20% of subjects enrolled in the study may have compensated cirrhosis]:
  - a) Cirrhosis is defined as any one of the following, below. Meeting any of these criteria will categorize the subject as cirrhotic.
    - i) Liver biopsy showing cirrhosis (e.g. Metavir score = 4 or Ishak score  $\geq 5$ )
    - ii) Fibroscan indicative of cirrhosis as evidenced by a result > 12.5 kPa
  - b) Absence of cirrhosis is defined as any one of the following:
    - i) Liver biopsy within 2 years prior to Screening showing absence of cirrhosis
    - ii) Fibroscan within 6 months prior to Baseline/Day 1 with a result of  $\leq 12.5$  kPa
- 9) Liver imaging within 6 months of Baseline/Day 1 to exclude hepatocellular carcinoma (HCC) is required in patients with cirrhosis
- 10) Screening ECG without clinically significant abnormalities
- 11) Subjects must have the following laboratory parameters at screening:
  - a) ALT  $\leq 10 \times$  the upper limit of normal (ULN)
  - b)  $AST \le 10 \times ULN$
  - c) Direct bilirubin  $\leq 1.5 \times ULN$
  - d) Platelets  $\geq 50,000/\mu L$
  - e)  $HbA_{1c} \le 8.5\%$
  - f) Creatinine clearance ( $CL_{cr}$ )  $\geq 50$  mL/min, as calculated by the Cockcroft-Gault equation {2202}
  - g) Hemoglobin  $\geq 11$  g/dL for female subjects;  $\geq 12$  g/dL for male subjects.
  - h) Albumin  $\geq 3g/dL$
  - i) INR  $\leq$  1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR.
- 12) Females of childbearing potential (as defined in Appendix 4) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Baseline/Day 1 prior to enrollment.

- 13) Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in Appendix 4.
- 14) Subject must be of generally good health, with the exception of chronic HCV infection, as determined by the Investigator.
- 15) Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

#### 4.3. Exclusion Criteria

Subjects who meet *any* of the following exclusion criteria are not to be enrolled in this study.

- 1) Current or prior history of any of the following:
  - a) Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
  - b) Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug.
  - c) Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
  - d) Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage).
  - e) Solid organ transplantation.
  - f) Significant pulmonary disease, significant cardiac disease or porphyria.
  - g) Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years. Subjects with psychiatric illness (without the prior mentioned conditions) that is well-controlled on a stable treatment regimen for at least 12 months prior to Baseline/Day 1 or has not required medication in the last 12 months may be enrolled.
  - h) Malignancy within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc.). Subjects under evaluation for possible malignancy are not eligible.
  - i) Significant drug allergy (such as anaphylaxis or hepatotoxicity).
- 2) If treatment-naïve, prior exposure to approved or experimental HCV-specific direct-acting antiviral agent(s). If treatment-experienced, prior exposure to approved or experimental HCV-specific direct-acting antiviral agent(s) other than NS3/4A protease inhibitors is prohibited.

- 3) Pregnant or nursing females.
- 4) Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, cholangitis).
- 5) Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
- 6) Donation or loss of more than 400 mL blood within 2 months prior to Baseline/Day 1.
- 7) Use of any prohibited concomitant medications as described in Section 5.4.
- 8) Administration of interferon or any HCV-directed treatment, other than the study drug, is prohibited from 12 weeks prior to Screening until completion of the final post-treatment follow-up visit.
- 9) Chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent > 10 mg/day), azathioprine or monoclonal antibodies such as infliximab.
- 10) Known hypersensitivity to SOF, LDV, or formulation excipients.

## 5. INVESTIGATIONAL MEDICINAL PRODUCTS

## **5.1.** Randomization and Treatment Codes

This is an open-label, non-randomized study. Every subject will receive SOF/LDV FDC tablet for 12 weeks. An Interactive Web Response System (IWRS) will be employed to manage subject enrollment and study drug dispensation.

## 5.2. Description and Handling of Sofosbuvir/Ledipasvir Fixed-Dose Combination

#### **5.2.1.** Formulation

Sofosbuvir (SOF)/ledipasvir (LDV) fixed-dose combination (FDC) tablets are orange, diamond-shaped, film-coated tablets containing 400 mg of SOF and 90 mg of LDV. The tablets are debossed with "GSI" on one side and "7985" on the other side. The SOF/LDV FDC tablets contain the following inactive ingredients: lactose monohydrate, copovidone, microcrystalline cellulose, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate, polyvinyl alcohol, titanium dioxide, talc, polyethylene glycol, FD&C yellow # 6 /sunset yellow FCF aluminum lake.

## 5.2.2. Packaging and Labeling

Sofosbuvir (SOF)/ledipasvir (LDV) fixed-dose combination (FDC) tablets are packaged in white, high density polyethylene (HDPE) bottles. Each bottle contains 30 tablets (Korea and Taiwan) or 28 tablets (China only) and a silica gel desiccant canister or sachet and polyester packing material. Each bottle is enclosed with a white, continuous thread, child-resistant screw cap with an induction-sealed, aluminum-faced liner.

All labels for SOF/LDV FDC bottles to be distributed to study centers in participating countries shall be labeled to meet all applicable requirements of the US Food and Drug Administration (FDA) and local regulations as applicable.

Sufficient quantities of SOF/LDV FDC tablets to complete the entire study will be shipped to the investigator or qualified designee from Gilead Sciences Materials & Logistics (or its designee).

# 5.2.3. Storage and Handling

Sofosbuvir (SOF)/ledipasvir (LDV) FDC bottles should be stored at controlled room temperature until required for administration. Controlled room temperature is defined as 25 °C; excursions are permitted between 15 °C and 30 °C.

All drug products should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability of the Investigational Medicinal Product (IMP) and to ensure proper product identification, the drug product should not be stored in a container other than the container in which they are supplied. Consideration should be given to handling, preparation, and

disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure through inhalation when handling SOF/LDV FDC.

## 5.3. Dosage and Administration of Sofosbuvir/Ledipasvir FDC

Sofosbuvir/Ledipasvir FDC tablet is to be administered once daily with or without food. Each subject must be given instructions to maintain approximately the same daily dosing interval between IMP doses. In order to maintain compliance with the treatment regimen, SOF/LDV FDC should be administered at approximately the same time each day.

For missed dose(s) of study medication, subjects should be instructed to take the missed dose(s) of IMP as soon as possible during the same day. Subjects should be cautioned never to double the next dose with a missed dose of IMP under any circumstances.

#### 5.4. Prior and Concomitant Medications

Concomitant medications taken within 30 days prior to Screening, up to and including the date of the visit four weeks after discontinuation of study treatment need to be recorded in the source documents and electronic case report form(s) (eCRFs).

Administration of interferon or any HCV-directed treatment, other than the study drug, is prohibited from 12 weeks prior to Screening until completion of the final post-treatment follow-up visit.

The following medications are prohibited during the screening period and for a minimum of 28 days prior to the Baseline/Day 1 visit through the end of treatment:

- Hematologic stimulating agents (e.g., erythropoiesis-stimulating agents (ESAs); granulocyte colony stimulating factor (GCSF); thrombopoietin (TPO mimetics)
- Chronic use of systemic immunosuppressants including, but not limited to, corticosteroids (prednisone equivalent of > 10 mg/day for > 2 weeks), azathioprine, or monoclonal antibodies (e.g., infliximab)
- Investigational agents or devices for any indication

Concomitant use of certain medications or herbal/natural supplements (inhibitors or inducers of drug transporters ie, P-gp) with study drug may result in pharmacokinetic interactions resulting in increases or decreases in exposure of study drug.

The use of amiodarone is prohibited from 60 days prior to Baseline/Day 1 through the end of treatment.

Examples of representative medications which are prohibited from 21 days prior to Baseline/Day 1 through the end of treatment are listed below:

Table 5-1. Disallowed and Concomitant Medications to be used with Caution

| Drug Class | Agents Disallowed | <b>Use with Caution</b> |
|---|---|---|
| Acid Reducing Agents <sup>a</sup> | | Proton- pump inhibitors, H2-<br>receptor antagonists, antacids |
| Anticonvulsants <sup>c</sup> | Phenobarbital, phenytoin, carbamazepine, oxcarbazepine | |
| Antimycobacterials <sup>c</sup> | Rifabutin, rifapentine, rifampin | |
| Cardiac Medications | Amiodarone <sup>e</sup> | Digoxin <sup>b</sup> |
| Herbal/Natural Supplements <sup>c</sup> | St. John's Wort, Echinacea, milk<br>thistle (ie, silymarin), Chinese herb<br>sho-saiko-to (or Xiao-Shai-Hu-<br>Tang) | |
| HMG-CoA Reductase Inhibitors <sup>d</sup> | Rosuvastatin | |

- a It is recommended to separate antacid and SOF/LDV FDC administration by 4 hours. H2-receptor antagonists may be administered simultaneously with or staggered from SOF/LDV FDC at a dose that does not exceed doses comparable to famotidine 40 mg twice daily. Proton-pump inhibitor doses comparable to omeprazole 20 mg can be administered simultaneously with SOF/LDV FDC. Proton-pump inhibitors should not be taken before SOF/LDV FDC.
- b Co-administration of SOF/LDV FDC with digoxin may increase the concentration of digoxin. Caution is warranted and therapeutic concentration monitoring of digoxin is recommended when co-administered with SOF/LDV FDC.
- c May result in a decrease in the concentrations of study drugs.
- d Use with study drug may result in an increase in the concentration of rosuvastatin, which is associated with increased risk of myopathy, including rhabdomyolysis.
- e May result in symptomatic bradycardia. Mechanism is not currently known. The use of amiodarone is prohibited from 60 days prior to Baseline/Day 1 through the end of treatment.

Medications for disease conditions **excluded** from the protocol (eg, HIV-1 infection, active cancer, transplantation) are not listed under this Concomitant Medication section and are disallowed in the study.

# 5.5. Accountability for SOF/LDV FDC

The investigator is responsible for ensuring adequate accountability of all used and unused IMP. This includes acknowledgement of receipt of each shipment of IMP (quantity and condition). All used and unused IMP dispensed to subjects must be returned to the site.

SOF/LDV FDC accountability records will be provided to each study site to:

- Record the date received and quantity of IMP kits.
- Record the date, subject number, subject initials, the IMP kit number dispensed.
- Record the date, quantity of used and unused IMP returned, along with the initials of the person recording the information.
Subjects must be instructed to bring back all bottles of study medication in the original container at <u>every post-baseline study visit</u> through the end of treatment.

Study medication will be reconciled using medication pill counts at every post-baseline visit by the investigator or designee (e.g., pharmacist, study coordinator) in order to monitor the subject's adherence with the medication regimen.

## 5.5.1. Investigational Medicinal Product Return or Disposal

Please refer to Section 9.1.7 for Investigational Medicinal Product Accountability and Return.

#### 6. STUDY PROCEDURES

Study visits will occur at Screening, Baseline/Day 1, and on-treatment at the end of Weeks 1, 2, 4, 6, 8, 10, and 12. All subjects will complete 4-week and 12-week Post-Treatment visits. In addition, all subjects with HCV RNA < LLOQ at the 12-week Post-Treatment visit will complete a 24-week Post-Treatment visit unless confirmed viral relapse occurs. The end of study will occur at the 12-week or 24-week Post-Treatment visit according to virologic response.

Administration of interferon or any HCV-directed treatment, other than the study drug, is prohibited from 12 weeks prior to Screening until completion of the final post-treatment follow-up visit.

The study procedures to be conducted for each subject enrolled in the study are presented in tabular form in Appendix 2 and described in the text that follows. Additional information is provided in the study procedures manual.

The investigator must document any deviation from protocol procedures and notify the sponsor or contract research organization (CRO).

Information on the specific laboratory parameters to be measured and clinical assessments to be performed are provided below.

## 6.1. Subject Enrollment and Treatment Assignment

#### **6.2.** Pretreatment Assessments

#### 6.2.1. Screening Visit (Day -28 to Day -1)

Screening assessments will be completed within 28 days of the Baseline/Day 1 visit. The screening window can be extended to 42 days for subjects requiring liver biopsy or additional HCV genotype testing.

Subjects will be screened to determine eligibility for participation in the study. The following will be performed and documented at screening:

- Obtain signed informed consent
  - A separate informed consent will be required from subjects participating in the intensive pharmacokinetic and/or pharmacogenomic sub-studies.
- Determine inclusion eligibility (Reference Section 4.2 and 4.3)
  - If the presence of cirrhosis is determined, then appropriate diagnostic imaging (e.g., CT or Ultrasound) should be performed to exclude the presence of hepatocellular carcinoma (HCC)

- Obtain medical history (Reference Section 6.6.2)
- Perform complete physical examination
- Obtain body height and weight
- Obtain vital signs (resting blood pressure, pulse, respiratory rate and temperature)
- Perform 12-lead ECG
- Assessment of AEs and concomitant medications
- Obtain blood samples for tests
  - Hematology & Chemistry
  - Coagulation tests
  - HCV RNA
  - Serum β-hCG pregnancy test for females of childbearing potential only
  - IL28B genotype
  - Determination of genotype and subtype of HCV infection
  - HCV antibody, HIV 1/2 antibody, and HBV surface antigen (HBsAg)
  - HbA1c
  - TSH
- Obtain urine sample for:
  - Urinalysis

Record any adverse events occurring after signing of the consent form.

Subjects meeting all of the inclusion criteria and none of the exclusion criteria will return to the clinic within 28-42 days after screening for entry into the study.

From the time of obtaining informed consent through the first administration of investigational medicinal product, record all serious adverse events (SAEs), as well as any non-serious adverse events related to protocol-mandated procedures on the adverse events case report form

(CRF/eCRF). All other untoward medical occurrences observed during the screening period, including exacerbation or changes in medical history are to be captured on the medical history CRF/eCRF. See Section 7 Adverse Events and Toxicity Management for additional details.

#### 6.3. Randomization

This is a non-randomized study. An Interactive Web Response System (IWRS) will be employed to manage subject enrollment and study drug dispensation.

#### 6.4. Treatment Assessments

#### 6.4.1. Baseline/Day 1 Visit

The following baseline tests and procedures must be completed prior to dosing/dispensing:

- Confirm eligibility
- Perform complete physical examination
- Obtain body weight
- Obtain vital signs
- Perform 12-lead ECG
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling
- Subject completes Health Related Quality of Life Survey, SF-36
- Obtain blood samples for:
  - Hematology & Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - Archive Sample (for subjects that have not opted out)
  - Pharmacogenomic testing (for subjects who have consented to participate in the Pharmacogenomic Substudy)

- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Drug Administration
  - Dispense study drugs as directed by the IWRS
  - Instruct the subject on the packaging, storage and administration of study drug
  - Instruct the subject on how to complete the subject diary
  - Observe the subject taking the first dose of study drugs and record the time of first dose.

## 6.4.2. Week 1 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 1.

- Obtain vital signs
- Perform 12-lead ECG
- Assessment of AEs and concomitant medications
- Obtain blood samples for:
  - Hematology & Chemistry
  - HCV RNA
  - Single PK Sample
  - Viral RNA Sequencing / Phenotyping Sample
- Complete medication pill count and review patient diary data with subject

## 6.4.3. Week 2 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 2:

- Obtain vital signs
- Assessment of AEs and concomitant medications
- Subject completes Health Related Quality of Life Survey, SF-36

- Obtain blood samples for:
  - Hematology & Chemistry
  - HCV RNA
  - Single PK Sample
  - Viral RNA Sequencing / Phenotyping Sample
  - If applicable at Week 2, collect serial PK substudy samples (for subjects who have consented to participate in the PK substudy)
- Complete medication pill count and review dosing diary data with subject

#### 6.4.4. Week 4 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 4:

- Obtain vital signs
- Assessment of AEs and concomitant medications
- Subject completes Health Related Quality of Life Survey, SF-36
- Obtain blood samples for:
  - Hematology & Chemistry
  - HCV RNA
  - Single PK Sample
  - Viral RNA Sequencing / Phenotyping Sample
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
  - If applicable at Week 4, collect serial PK substudy samples (for subjects who have consented to participate in the PK substudy)
- Complete medication pill count and review patient diary data with subject
- Dispense study drugs as directed by the IWRS

#### 6.4.5. Week $6 (\pm 3 \text{ days})$

The following procedures/assessments are to be completed at the end of Week 6.

- Obtain vital signs
- Assessment of AEs and concomitant medications
- Obtain blood samples for:
  - Hematology & Chemistry
  - HCV RNA
  - Single PK Sample
  - Viral RNA Sequencing / Phenotyping Sample
- Complete medication pill count and review patient diary data with subject

#### 6.4.6. Week 8 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 8:

- Obtain vital signs
- Assessment of AEs and concomitant medications
- Subject completes Health Related Quality of Life Survey, SF-36
- Obtain blood samples for:
  - Hematology & Chemistry
  - HCV RNA
  - Single PK Sample
  - Viral RNA Sequencing / Phenotyping Sample
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Complete medication pill count and review patient diary data with subject
- Dispense study drugs as directed by the IWRS

## 6.4.7. Week $10 (\pm 3 \text{ days})$

The following procedures/assessments are to be completed at the end of Week 10.

- Obtain vital signs
- Assessment of AEs and concomitant medications
- Obtain blood samples for:
  - Hematology & Chemistry
  - HCV RNA
  - Single PK Sample
  - Viral RNA Sequencing / Phenotyping Sample
- Complete medication pill count and review patient diary data with subject

## 6.4.8. Week 12 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 12:

- Perform complete physical examination
- Obtain body weight
- Obtain vital signs
- Perform 12-lead ECG
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling
- Subject completes Health Related Quality of Life Survey, SF-36
- Obtain blood samples for:
  - Hematology & Chemistry
  - Coagulation tests
  - HCV RNA
  - Single PK Sample

- Viral RNA Sequencing / Phenotyping Sample
- Archive Sample (for subjects that have not opted out)
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Complete medication pill count and review patient diary data with subject

### 6.4.9. Early Termination (ET)/Unscheduled Visit

A subject should attend an unscheduled visit if requested by the sponsor or the investigator. The assessments at the unscheduled visits are at the investigator's discretion. At all unscheduled visits initiated for the purpose of confirming virologic failure, a Viral RNA Sequencing / Phenotyping Sample must be collected.

The Sponsor (e.g. Medical Monitor and Clinical Program Manager)/ CRO must be informed, as soon as possible, when a subject prematurely discontinues treatment. The primary reason for premature treatment discontinuation must be provided to the Sponsor/ CRO.

If a subject discontinues treatment early for any reason then the following assessments for the Early Termination (ET) Visit must be performed:

- Perform complete physical examination
- Obtain body weight
- Obtain vital signs
- Perform 12-lead ECG
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling
- Subject completes a Health Related Quality of Life Survey, SF-36
- Obtain blood samples for:
  - Hematology & Chemistry
  - Coagulation tests
  - HCV RNA

- Single PK Sample
- Viral RNA Sequencing / Phenotyping Sample
- Archive Sample (for subjects that have not opted out)
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Complete medication pill count and review dosing diary data with subject

#### 6.5. Post-Treatment Assessments

All subjects must complete the Post-Treatment Week 4 and Week 12 visits. For subjects who have completed an ET visit, the post-treatment Week 4 and Week 12 follow-up visits will be scheduled at 4 and 12 weeks after the last dose of study drug. All subjects with HCV RNA < LLOQ at the 12-week Post-Treatment visit will also complete the 24-week Post-Treatment visit, unless viral relapse is determined.

#### 6.5.1. Post Treatment Week 4 (± 5 days)

The following procedures/assessments are to be completed for all subjects, 4 Weeks after taking the last dose of study drug:

- Obtain vital signs
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling
- Subject completes a Health Related Quality of Life Survey, SF-36
- Obtain blood samples for:
  - Hematology & Chemistry
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only

All subjects, including those who prematurely discontinue study drug, must return for Post Treatment Visit at Week 12.

## 6.5.2. Post Treatment Weeks 12 and 24 ( $\pm$ 5 days)

The following procedures/assessments are to be completed for the Post-treatment Week 12 and 24 Visits:

- Obtain body weight
- Obtain vital signs
- Subject completes a Health Related Quality of Life Survey, SF-36 (Post treatment Week 12 only)
- Obtain blood samples for:
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample

Subjects with HCV RNA < LLOQ at the Post-Treatment Week 12 Visit will return at the post-treatment Week 24 Visit.

#### 6.6. Procedures and Specifications

## 6.6.1. Clinical Laboratory Analytes

<u>Hematology:</u> Hematocrit, Hemoglobin (Hb), Platelet count, Red blood cell count (RBC), White blood cell count (WBC) with differential (absolute and percentage) including Lymphocytes, Monocytes, Neutrophils, Eosinophils, Basophils, Reticulocyte count and MCV.

Coagulation: INR, Prothrombin time (PT), Activated partial thromboplastin time (APTT).

<u>Chemistry:</u> Alanine aminotransferase (ALT/SGPT), Aspartate aminotransferase (AST/SGOT), Albumin, Alkaline phosphatase, Creatinine, Total Bilirubin (reflex to Direct Bilirubin), Direct Bilirubin at Screening only, Glucose, Lipase, Potassium, Sodium; Gamma-glutamyl transferase (GGT) at Baseline only.

<u>Urinalysis:</u> Appearance, Blood, Color, Glucose, Leukocyte esterase, pH, Protein, Urobilinogen. Reflex to microscopic urinalysis if dipstick result is abnormal.

<u>Virological Tests</u>: Serologies for HCV, HBV and HIV. HCV RNA will be measured using the COBAS<sup>®</sup> TaqMan<sup>®</sup> HCV Test, v2.0 for Use with the High Pure System or COBAS<sup>®</sup> AmpliPrep / COBAS<sup>®</sup> TaqMan<sup>®</sup> HCV Test, v2.0. HCV genotype and subtype will be determined using the Siemens VERSANT<sup>®</sup> HCV Genotype INNO-LiPA 2.0 Assay. Gilead reserves the right to use alternate assays for HCV RNA and HCV genotype should the above assays become unavailable or are not definitive.

IL28B genotype will be determined by polymerase chain reaction (PCR) amplification of the SNP, rs12979860, with sequence specific forward and reverse primers and allele specific

fluorescently labeled TaqMan® MGB probes. Gilead reserves the rights to use an alternate assay for IL28B determination should the above assay become unavailable.

<u>Pregnancy Tests</u>: Serum β-hCG or Urine β-hCG (if positive, requires immediate confirmation with Serum β-hCG)

Additional Tests: Hemoglobin A1c (HbA1c), and TSH (reflex free T4).

#### 6.6.2. Medical History

Medical history including details regarding illnesses and allergies, date(s) of onset, and whether condition(s) is currently ongoing, and medication history will be collected on all subjects during screening. Additionally, for treatment naïve subjects, any relative or absolute contraindications to interferon treatment ("IFN ineligible") should be identified. Information related to HCV infection will also be collected.

For treatment-experienced subjects, obtain HCV treatment history, in order to categorize the patient as either IFN-intolerant, non-responder or relapse/breakthrough, defined as:

- IFN-intolerant: Subjects considered to be IFN-intolerant must (according to investigator judgment) have sufficiently recovered from IFN-related clinical adverse events and/or laboratory abnormalities prior to Screening. In addition, all other protocol eligibility criteria must be met.
- Non-Responder: Subject did not achieve undetectable HCV RNA levels (HCV RNA ≥ LLOQ) while on treatment. For Peg-IFNα/IFN/RBV non-responders, subjects should be further defined as Null or Partial Responders:
  - Null Responders: HCV RNA < 2 Log10 reduction during the first 12 weeks of treatment.
  - Partial Responders: HCV RNA ≥ 2 Log10 reduction during the first 12 weeks of treatment.
- Relapse/Breakthrough: Subject achieved undetectable HCV RNA levels (HCV RNA < LLOQ) during treatment or within 4 weeks of end of treatment, but did not achieve a sustained virologic response (SVR).

# **6.6.3.** Complete Physical Examination

A complete physical examination must include source documentation of general appearance, and the following body systems: Head, neck and thyroid; eyes, ears, nose, throat, mouth and tongue; chest (excluding breasts); respiratory; cardiovascular; lymph nodes, abdomen; skin, hair, nails; musculoskeletal; neurological.

## 6.6.4. Vital Signs

Assessment of vital signs will include measurement of resting blood pressure, pulse, respiratory rate, and temperature.

Blood pressure will be measured using the following standardized process:

- Subject should sit for  $\geq 5$  minutes with feet flat on the floor and measurement arm supported so that the midpoint of the manometer cuff is at heart level;
- Use a mercury sphygmomanometer or automatic blood pressure device with an appropriately sized cuff with the bladder centered over the brachial artery;
- Measure and record the blood pressure to the nearest 2 mmHg mark on the manometer or to the nearest whole number on an automatic device.

#### 6.6.5. Creatinine Clearance

Creatinine clearance is calculated by the Cockcroft-Gault equation {2202} using actual body weight (BW).

Male: 
$$CL_{cr} (mL/min) = [\underline{140 - age (years)}] \times \underline{BW(kg)}$$

Female: 
$$CL_{cr} (mL/min) = \underline{[140 - age (years)] \times BW(kg) \times 0.85}$$
  
 $72 \times S_{cr}$ 

 $S_{cr}$  = serum creatinine (mg/dL)

#### 6.6.6. 12-Lead ECGs

Subjects will be required to rest in a supine position for  $\geq 5$  minutes prior to making a recording.

The investigator (or qualified designee) should review the ECG traces recorded in real time for clinically significant abnormalities. On-treatment ECGs should be compared to the subject's Baseline as part of routine safety monitoring.

# 6.6.7. Viral RNA Sequencing / Phenotyping Sample

Plasma samples will be collected at Baseline/Day 1 and each additional visit for viral sequence analysis. At any unscheduled visit initiated for the purpose of confirming virologic breakthrough, a plasma sample for viral sequence analysis must be collected. Untested samples may be archived

Details regarding the collection, processing, and shipping of samples will be included in the lab manual.





## 6.6.9. Single Pharmacokinetic (PK) Sample

Single PK blood samples will be collected for all subjects at each on-treatment visit after Baseline/Day 1 and archived for PK analysis of SOF (and its metabolites GS-566500 and GS-331007) and LDV.

Details regarding the collection, processing, and shipping of samples will be included in the lab manual.





# 6.6.11. Pharmacogenomic (PG) Substudy

PPD



## 6.6.12. Pregnancy Testing

All females of childbearing potential will have urine pregnancy testing every 4 weeks during the dosing period and for a minimum of 1 month following the last dose of study drug. In the event of a positive urine pregnancy test result, subjects will be instructed to stop study drugs immediately and return to the clinic as soon as possible for a confirmatory serum pregnancy test.

#### 6.6.13. Health Related Quality of Life Survey

A health related quality of life survey, SF-36 will be completed by patients at Baseline/Day 1, On-treatment Weeks 2, 4, 8, 12, Post-treatment Weeks 4 and 12, and Early Termination (if applicable). The subject should read the questionnaire by himself/herself and write/mark answers directly onto the questionnaire.

#### 6.7. Assessments for Premature Discontinuation from Study

If a subject discontinues study dosing (for example, as a result of an AE), every attempt should be made to keep the subject in the study and continue to perform the required study-related follow-up and procedures (see Section 6.4.9). If this is not possible or acceptable to the subject or investigator, the subject may be withdrawn from the study.

#### 7. ADVERSE EVENTS AND TOXICITY MANAGEMENT

# 7.1. Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events

#### 7.1.1. Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also include pre- or post treatment complications that occur as a result of protocol specified procedures, lack of efficacy, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increase in severity or change in nature during or as a consequence of participation in the clinical study will also be considered AEs.

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an adverse event and must be reported.
- Pre-existing diseases, conditions, or laboratory abnormalities present or detected before the screening visit that do not worsen
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions)
- Overdose without clinical sequelae (see Section 7.7.1)
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be pre-existing and should be documented on the medical history CRF.

#### 7.1.2. Serious Adverse Events

A **serious adverse event** (SAE) is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)
- In-patient hospitalization or prolongation of existing hospitalization

- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse. For the avoidance of doubt, infections resulting from contaminated medicinal product will be considered a medically important event and subject to expedited reporting requirements.

#### 7.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified sub-investigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

#### 7.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to IMP therapy using clinical judgment and the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the IMP. For SAEs, an alternative causality must be provided (eg, pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).
- Yes: There is reasonable possibility that the event may have been caused by the investigational medicinal product.

It should be emphasized that ineffective treatment should not be considered as causally related in the context of adverse event reporting.

The relationship to study procedures (eg, invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the study procedure.
- Yes: The adverse event occurred as a result of protocol procedures, (eg., venipuncture)

# 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events to Gilead or CRO

All SAEs, regardless of causal relationship, that occur after the subject first consents to participate in the study (ie, signing the informed consent) and throughout the duration of the study, including the protocol-required post treatment follow-up period, must be reported to the CRF/eCRF database and Gilead Drug Safety and Public Health (DSPH) as instructed. This also includes any SAEs resulting from protocol-mandated procedures performed from screening onwards.

All AEs, regardless of causal relationship, that occur from initiation of study medication until 4 weeks after last administration of study IMP must be reported to the CRF/eCRF database as instructed.

All AEs should be followed up until resolution or until the adverse event is stable, if possible. Gilead Sciences may request that certain AEs be followed beyond the post-treatment follow up period.

Investigators are not obligated to actively seek SAEs after post treatment follow-up. However, if the investigator learns of any SAEs that occur after study participation has concluded, i.e., after the 12-week or 24-week post treatment visit (as applicable) and the event is deemed relevant to the use of IMP, he/she should promptly document and report the event to Gilead DSPH. Gilead DSPH contact information is as follows: Email: Safety\_FC@gilead.com and Fax: +1 (650) 522-5477.

• All AEs and SAEs will be recorded in the CRF/eCRF database within the timelines outlined in the CRF/eCRF completion guideline.

#### Electronic Serious Adverse Event (eSAE) Reporting Process

- Site personnel record all SAE data in the eCRF database and from there transmit the SAE information to Gilead DSPH within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.
- If for any reason it is not possible to record the SAE information electronically, ie, the eCRF database is not functioning, record the SAE on the paper serious adverse event reporting form and submit within 24 hours as described above.
  - As soon as it is possible to do so, any SAE reported via paper must be transcribed into the eCRF Database according to instructions in the eCRF completion guidelines.
  - If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.

CRO and Gilead Sciences Pharmacovigilance Representative contact information is as follows:

CRO Pharmacovigilance SAE Hotline: + 65 6221 8582
Representative Korea: + 00308 13 2766
(for sites in Korea and Taiwan): Taiwan: + 00801 10 4423

E-mail: medical\_singapore@parexel.com

CRO Pharmacovigilance China: Quintiles

Representative E-mail: PhV Gilead@quintiles.com

(for sites in China):

CRO Medical Monitor Name: Viola Yang

(for sites in Korea and Taiwan): Phone: PPD

Fax: PPD E-mail: PPD

CRO Medical Monitor Name: Ian Escudero

(for sites in China) Phone: PPD

Fax: PPD E-mail: PPD

Gilead Sciences Medical Monitor Name: Chohee Yun MD

(Back-Up): Phone: PPD Fax: PPD

E-mail: PPD

- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and other
  documents are also to be submitted by e-mail or fax when requested and applicable.
   Transmission of such documents should occur without personal subject identification,
  maintaining the traceability of a document to the subject identifiers.
- Additional information may be requested to ensure the timely completion of accurate safety reports.

Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's CRF/eCRF and the event description section of the SAE form.

# 7.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the EU Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory

agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports. The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

# 7.5. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to IMP interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 7.1.1. and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

Severity should be recorded and graded according to the GSI Grading Scale for Severity of AEs and Laboratory Abnormalities (Appendix 3). For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

#### 7.6. Subject Stopping Rules

The Medical Monitor must be consulted prior to dose discontinuation of SOF/LDV FDC unless the investigator believes that immediate action is warranted to ensure the continued safety of the subject.

Due to a clinical or laboratory event, administration of study drug may be discontinued. There is no option for SOF/LDV FDC dose reduction. If SOF/LDV FDC is stopped due to toxicity, it must not be restarted; if SOF/LDV FDC is discontinued, the subject must complete an ET visit. Post-treatment 4-Week and 12-Week visits must also be scheduled, 4 and 12 weeks from the last dose of study drug. Subjects with HCV RNA < LLOQ at the 12-week Post-Treatment visit will complete the 24-week Post-Treatment visit, unless viral relapse is determined.

Subjects who meet any of the following laboratory criteria must stop study medication:

- Elevation of ALT and/or AST > 5x Baseline/Day 1 or nadir, confirmed by immediate repeat testing
- Abnormal elevation of ALT > 3 x Baseline/Day 1 *and* total bilirubin > 2 x ULN, confirmed by immediate repeat testing

- Elevation of ALT  $\geq$  15 x ULN, confirmed by immediate repeat testing
- Any Grade 3 or greater rash associated with constitutional symptoms
- Any Grade 4 adverse event or laboratory abnormality assessed as related to SOF/LDV FDC

#### 7.7. Special Situations Reports

#### 7.7.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, and pregnancy reports regardless of an associated AE. Also includes reports of adverse reactions in infants following exposure from breastfeeding, and reports of adverse reactions associated with product complaints and reports arising from occupational exposure.

A pregnancy report is used to report any pregnancy following maternal or paternal exposure to the medicinal product.

Medication error is any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in the control of the health care provider, subject, or consumer.

Abuse is defined as persistent or sporadic intentional excessive use of a medicinal product by a subject.

Misuse is defined as any intentional and inappropriate use of a medicinal product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of a medicinal product given per administration or cumulatively which is above the maximum recommended dose as per protocol. In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Product complaint is defined as complaints arising from potential deviations in the manufacture, packaging, or distribution of the medicinal product.

## 7.7.2. Instructions for Reporting Special Situations

## 7.7.2.1. Instructions for Reporting Pregnancies

The investigator should report all pregnancies that are identified after the subject first consents to participate in the study (ie, signs the informed consent) and throughout the study, including the post study drug follow-up period, to the CRO Pharmacovigilance Representative using the pregnancy report form within 24 hours of becoming aware of the pregnancy.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in the Serious Adverse Events section (Section 7.3). Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported to the CRO Pharmacovigilance Representative.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to the CRO Pharmacovigilance Representative using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH. Gilead DSPH contact information is as follows: Email: Safety FC@gilead.com and Fax: +1 (650) 522-5477.

Pregnancies of female partners of male study subjects exposed to Gilead study drugs must also be reported and relevant information should be submitted to the CRO Pharmacovigilance Representative using the pregnancy and pregnancy outcome forms within 24 hours. Monitoring of the subject's partner should continue until the conclusion of the pregnancy. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH, fax number +1 650 522-5477 or email Safety FC@gilead.com.

Refer to Appendix 4 for Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements.

# 7.7.2.2. Reporting Other Special Situations

All other special situation reports must be reported on the special situations report form and forwarded to the CRO Pharmacovigilance Representative within 24 hours of the investigator becoming aware of the situation. These reports must consist of situations that involve study IMP, but do not apply to concomitant medications. Except for situations that result in AEs, special situations involving concomitant medications will not be reported. Any inappropriate use of medications prohibited by this protocol should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE CRF/eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome will be reported, when available.

#### 8. STATISTICAL CONSIDERATIONS

## 8.1. Analysis Objectives and Endpoints

#### 8.1.1. Analysis Objectives

The primary analysis objectives of this study are:

- To determine the antiviral efficacy of combination treatment with sofosbuvir (SOF)/ledipasvir (LDV) fixed-dose combination (FDC) as measured by the proportion of subjects with sustained virologic response (SVR) 12 weeks after discontinuation of therapy (SVR12, defined as HCV RNA < lower limit of quantitation [LLOQ] 12 weeks post treatment).
- To evaluate the safety and tolerability of SOF/LDV FDC as assessed by review of the accumulated safety data

The secondary objectives of this study are as follows:

- To determine the proportion of subjects who attain SVR at 4 and 24 weeks after discontinuation of therapy (SVR4 and SVR24)
- To evaluate the kinetics of circulating HCV RNA during treatment and after treatment discontinuation
- To evaluate the emergence of viral resistance to SOF and LDV during treatment and after treatment discontinuation

The exploratory objectives of this study are:



#### 8.1.2. Primary Endpoint

The primary efficacy endpoint is SVR12 (HCV RNA <LLOQ 12 weeks after discontinuation of therapy) in the Full Analysis Set (FAS) population.

The primary safety endpoint is any AE leading to permanent discontinuation of study drug.

## 8.1.3. Secondary Endpoint

Secondary efficacy endpoints include the proportion of subjects with: HCV RNA < LLOQ at 4 and 24 weeks after discontinuation of therapy (SVR4 and SVR24); viral breakthrough; relapse; and HCV RNA change from baseline.

#### 8.1.4. Other Endpoints of Interest

Additional efficacy evaluations may include ALT normalization; and the health related quality of life endpoints.

#### 8.2. Analysis Conventions

All individual subject data will be listed as measured. All statistical summaries and analyses will be performed using SAS® software (SAS Institute, Cary, North Carolina, USA).

Last dose of study drug refers to the last dose of SOF/LDV FDC and will be used in the definition of treatment-emergent AEs and laboratory abnormalities as well as the efficacy endpoints of SVR at various post-treatment time points.

## 8.2.1. Analysis Sets

#### 8.2.1.1. Efficacy

The analysis set for antiviral activity analyses will be the Full Analysis Set (FAS) which includes subjects who were enrolled and received at least one dose of study drug and have chronic genotype (1a, 1b, or mixed 1a/1b) HCV infection.

#### 8.2.1.2. Safety

The primary analysis set for safety analyses is defined as subjects who were enrolled and received at least one dose of study drug.

Treatment-emergent data will be analyzed and defined as data collected from the first dose of study drug through the date of the last dose of study drug plus 30 days.

#### 8.2.1.3. Pharmacokinetics

The PK analysis set will include all subjects who are enrolled and have received at least one dose of study drug and for whom concentration data of analytes [SOF, LDV, and metabolite(s), as appropriate] are available. The PK analysis set will be used for analyses of general PK.

## 8.3. Data Handling Conventions

Missing data can have an impact upon the interpretation of the trial data. In general, values for missing data will not be imputed.

For the analysis of post-baseline categorical efficacy endpoints, if a data point is missing and is immediately preceded and followed in time by values that are deemed successes, then the missing data point will be termed a success; otherwise the data point will be termed a failure.

Any subject with missing data due to premature discontinuation of the study will be considered a failure at the time points on, or following, the date of discontinuation. If no HCV RNA values are obtained after the last dose of study medication, the subject will be considered a treatment failure for the SVR endpoints.

Where appropriate, safety data for subjects that did not complete the study will be included in summary statistics. For example,

- If a subject received study medication, the subject will be included in a summary of adverse events according to the treatment received; otherwise, if the subject is not dosed then they will be excluded from the summary.
- If safety laboratory results for a subject are missing for any reason at a time point, the subject will be excluded from the calculation of summary statistics for that time point. If the subject is missing a pre-dose value, then the subject will be excluded from the calculation of summary statistics for the pre-dose value and the change from pre-dose values.

Values for missing safety laboratory data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available. If no pre-treatment laboratory value is available, the baseline value will be assumed to be normal (i.e., no grade [Grade 0]) for the summary of graded laboratory abnormalities.

Values for missing vital signs data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available.

HCV RNA values below the LLOQ for the assay will be set to the lower limit minus 1 for calculation of summary statistics for the actual HCV RNA values and the change from baseline values by study visit. The reported values will be provided in the HCV RNA listing.

For selected analyses of early time point data, HCV RNA data (IU/mL) may be transformed to the logarithmic (base 10) scale (log<sub>10</sub> IU/mL).

PK concentration values below the lower limit of quantitation (BLQ) will be treated as zero for determination of summary and order statistics. Individual values that are BLQ will be presented as "BLQ" in the concentration data listing. For the presentation of summary and order statistics, if at least 1 subject has a concentration value BLQ for the time point, then the minimum value will be displayed as "BLQ". If more than 50% of the subjects have a concentration data value

BLQ for the time point, then the minimum and median values will be displayed as "BLQ". If all subjects have concentration data values BLQ for the time point, then all order statistics (minimum, first quartile [Q1], median, third quartile [Q3], maximum) will be displayed as "BLQ".

Exposure parameters that are selected for statistical analysis will be natural log-transformed. Concentration values that are BLQ will be excluded for any ratio or natural log-transformed statistical analysis.

#### 8.3.1. Interim Analysis

An interim analysis will be performed after all subjects enrolled from Korea and Taiwan have been followed through 12 weeks post-treatment or discontinued from the study to support regulatory submissions in these two countries.

# 8.4. Demographic Data and Baseline Characteristics

Demographic and baseline measurements will be summarized using standard descriptive methods by treatment-naive and treatment-experienced subjects.

Demographic summaries will include sex, self-identified race/ethnicity, and age.

Baseline characteristic data will include a summary of body mass index, HCV RNA level (log<sub>10</sub> IU/mL), HCV genotype (1a or 1b, or mixed 1a/1b), IL28B genotype, presence/absence of cirrhosis, baseline ALT level, and additional endpoints as necessary.

#### 8.5. Efficacy Analysis

#### 8.5.1. Primary Analysis

The primary efficacy endpoint is SVR12 (HCV RNA <LLOQ 12 weeks after discontinuation of therapy) in the FAS population. The primary analysis will be performed after all enrolled subjects have been followed through 12 weeks post-treatment or discontinued from study.

The primary efficacy analysis described below will compare the observed SVR12 rate for the investigational regimen (i.e., SOF/LDV FDC for 12 weeks) versus the historical SVR null rate in treatment—naïve Korean subjects and in treatment—naïve Chinese subjects, respectively.

In addition, a point estimate with a two-sided 95% exact confidence interval using the binomial distribution (Clopper-Pearson method) {20839} will be constructed for the SVR12 rate by treatment-naïve and treatment-experienced subjects for each region (i.e., China, Korea or Taiwan), Korea plus Taiwan and overall (i.e., China plus Korea plus Taiwan).

#### **Treatment-Naïve Subjects**

In the primary efficacy analysis the SVR12 rate from Korea and China will be compared to the adjusted historical SVR null rate of 49% in Korea and historical control rate of 57% in China, respectively (as calculated in Appendix 5) using a two-sided exact one-sample binomial test.

The hypothesis for superiority in Korea is:

- H0: SVR12 rate = 49%,
- H1: SVR12 rate  $\neq$  49%.

The hypothesis for superiority in China is:

- H0: SVR12 rate = 57%,
- H1: SVR12 rate ≠ 57%.

#### **Treatment-Experienced Subjects**

There is no treatment option available in China, Korea or Taiwan for treatment-experienced patients with GT-1 infection. In the absence of effective antiviral therapy, spontaneous clearance of the HCV is rare. Consequently a nominal SVR rate of 5% is assumed for treatment-experienced subjects.

No statistical hypothesis testing will be performed in treatment-experienced subjects. For each region (i.e., China, Korea or Taiwan), Korea plus Taiwan, and overall (i.e., China plus Korea plus Taiwan), a point-estimate with two-sided 95% exact confidence interval using the binomial distribution (Clopper-Pearson method) will be constructed for the SVR12 rate.

### 8.5.2. Secondary Analysis

The proportion of subjects with HCV RNA below LLOQ over time (including SVR12) will be presented by treatment-naive and treatment-experienced subjects for each region (i.e., China, Korea or Taiwan), Korea plus Taiwan, and overall (i.e., China plus Korea plus Taiwan) in tabular and graphical form.

Descriptive summaries and listings will be provided for additional efficacy evaluations including the proportion of subjects who experience virologic failure, ALT normalization, serum HCV RNA actual values and change from baseline and health related quality of life endpoints.



Details on efficacy analyses will be described in the statistical analysis plan.

# 8.6. Safety Analysis

Safety will be evaluated by assessment of clinical laboratory tests, physical examinations, vital signs measurements, at various time points during the study, and by the documentation of AEs.

All safety data collected on or after the first dose of study drug administration up to 30 days after the last dose of study drug will be summarized for each region (i.e., China, Korea or Taiwan), Korea plus Taiwan, and overall (i.e., China plus Korea plus Taiwan). Safety endpoints will be summarized as the number (proportion) of subjects with events or abnormalities for categorical data or as an 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data.

#### 8.6.1. Extent of Exposure

A subject's extent of exposure to IMP data will be generated from the IMP administration data. Exposure data will be summarized.

#### **8.6.2.** Adverse Events

Clinical and laboratory adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database.

Events will be summarized on the basis of the date of onset for the event. A treatment-emergent adverse event will be defined as any new or worsening adverse event that begins on or after the date of first dose of IMP up to the date of last dose of IMP plus 30 days.

Summaries (number and percentage of subjects) of treatment-emergent adverse events (by SOC, HLT, and PT) will be provided:

- All AEs,
- All study drug-related AEs,
- Combined Grade 2, 3 and 4 AEs,
- Combined Grade 3 and 4 AEs,
- Combined Grade 2, 3 and 4 study drug-related AEs,
- Combined Grade 3 and 4 study drug-related AEs,
- All AEs that caused permanent discontinuation from study drug,
- All AEs that caused change in dose or temporary interruption of study drug,

- All SAEs (including death), and
- All study drug-related SAEs

All AEs collected during the course of the study will be presented in data listings.

#### **8.6.3.** Laboratory Evaluations

Selected laboratory data (n, mean, SD, median, Q1, Q3, minimum, and maximum) will be summarized at study visits along with corresponding change from baseline.

Graded laboratory abnormalities will be defined using the laboratory toxicity grading scheme defined in Appendix 3 of this protocol. The incidence of treatment-emergent laboratory abnormalities, defined as values that increase by at least one toxicity grade from baseline at any time post-baseline up to the date of last dose of study drug plus 30 days will be summarized. If baseline data are missing, then any post-baseline graded abnormality (i.e., at least Grade 1) will be considered treatment emergent.

All laboratory abnormalities will be included in the listings of laboratory data.

## 8.7. Pharmacokinetic Analysis

. Intensive plasma concentrations of the study drug and metabolite(s) over time, if analyzed, will be summarized using descriptive statistics. Details of the analysis plan will be provided in the statistical analysis plan. Population PK parameters for the study drugs and metabolite(s), as applicable, will be estimated and summarized using descriptive statistics

#### 8.8. Sample Size

#### **Treatment-Naïve Subjects:**

A sample size of 40 Korean subjects in the treatment-naïve group will provide at least 90% power to detect a 27% improvement in SVR12 rate from the adjusted historical control rate of 49% using 2-sided exact one-sample binomial test at significant level of 0.05.

A sample size of 100 Chinese subjects in the treatment-naïve group will provide at least 90% power to detect a 17% improvement in SVR12 rate from the historical control rate of 57% using 2-sided exact one-sample binomial test at significant level of 0.05.

In addition, with 40 subjects in Korea (or Taiwan), the 2 sided 95% exact confidence interval will extend at most 32% in length. With 80 subjects (Korea plus Taiwan) in the treatment-naive group a two-sided 95% exact confidence interval will extend at most 23% in length. With 100 subjects in China, the 2 sided 95% exact confidence interval for the SVR12 rate will extend at most 20% in length.

## **Treatment-Experienced Subjects:**

For Treatment Experienced subjects, a confidence interval approach will be used to justify the sample size given that our goal is to characterize the SVR rate in a population with limited treatment options and not to test a specific hypothesis. With 40 subjects in Korea (or Taiwan), the 2 sided 95% exact confidence interval will extend at most 32% in length. With 80 subjects (Korea plus Taiwan) in the treatment-experienced group, a two-sided 95% exact confidence interval will extend at most 23% in length. With 100 subjects in China, the 2 sided 95% exact confidence interval for the SVR12 rate will extend at most 20% in length.

## 9. **RESPONSIBILITIES**

## 9.1. Investigator Responsibilities

#### 9.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki (as amended in Edinburgh, Tokyo, Venice, Hong Kong, and South Africa), International Conference on Harmonisation (ICH) guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject. These standards are consistent with the European Union Clinical Trials Directive 2001/20/EC and Good Clinical Practice Directive 2005/28/EC.

The investigator will ensure adherence to the basic principles of Good Clinical Practice, as outlined in 21 CFR 312, subpart D, "Responsibilities of Sponsors and Investigators," 21 CFR, part 50, 1998, and 21 CFR, part 56, 1998.

The investigator and all applicable subinvestigators will comply with 21 CFR, Part 54, 1998, providing documentation of their financial interest or arrangements with Gilead, or proprietary interests in the investigational drug under study. This documentation must be provided prior to the investigator's (and any subinvestigator's) participation in the study. The investigator and subinvestigator agree to notify Gilead of any change in reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date when the last subject completes the protocol-defined activities.

This study is also subject to and will be conducted in accordance with 21 CFR, part 320, 1993, "Retention of Bioavailability and Bioequivalence Testing Samples."

# 9.1.2. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) Review and Approval

The investigator (or sponsor as appropriate according to local regulations) will submit this protocol, informed consent form, and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) to an IRB/IEC. The investigator will not begin any study subject activities until approval from the ECIRB/IEC and/or Regulatory Body has been documented and provided as a letter to the investigator.

Before implementation, the investigator will submit to and receive documented approval from the ECIRB/IEC and/or Regulatory Body IRB/IEC any modifications made to the protocol or any accompanying material to be provided to the subject after initial IRB/IEC approval, with the exception of those necessary to reduce immediate risk to study subjects.

#### 9.1.3. Informed Consent

The investigator is responsible for obtaining written informed consent from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. The investigator must use the most current IRB- or IEC-approved informed consent form (ICF) for documenting written informed consent. Each informed consent (or assent as applicable) will be appropriately signed and dated by the subject or the subject's legally authorized representative and the person conducting the consent discussion, and also by an impartial witness if required by IRB or IEC or local requirements. PPD

. The

Pharmacogenomic consent form will inform subjects about pharmacogenomic testing and sample retention, and their right to receive clinically relevant pharmacogenomic analysis results.

#### 9.1.4. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject initials, date of birth, another unique identifier (as allowed by local law) and an identification code will be recorded on any form or biological sample submitted to the Sponsor, IRB [or] IEC, or laboratory. Laboratory specimens must be labeled in such as way as to protect subject identity while allowing the results to be recorded to the proper subject. Refer to specific laboratory instructions. NOTE: The investigator must keep a screening log showing codes, names, and addresses for all subjects screened and for all subjects enrolled in the trial. Subject data will be processed in accordance with all applicable regulations.

The investigator agrees that all information received from Gilead, including but not limited to the investigator brochure, this protocol, CRF/eCRF, the IMP, and any other study information, remain the sole and exclusive property of Gilead during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

#### 9.1.5. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following two categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, CRF and query forms, IRB [or] IEC and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include sequential notes containing at least the following information for each subject:

- Subject identification (name, date of birth, gender);
- Documentation that subject meets eligibility criteria, ie, history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria);
- Documentation of the reason(s) a consented subject is not enrolled
- Participation in study (including study number);
- Study discussed and date of informed consent;
- Dates of all visits;
- Documentation that protocol specific procedures were performed;
- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of IMP, including dates of dispensing and return;
- Record of all adverse events and other safety parameters (start and end date, and including causality and severity);
- Concomitant medication (including start and end date, dose if relevant; dose changes);
- Date of study completion and reason for early discontinuation, if it occurs.

All clinical study documents must be retained by the investigator until at least 2 years or according to local laws, whichever is longer, after the last approval of a marketing application in an ICH region (ie, United States, Europe, or Japan) and until there are no pending or planned marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if specified by regulatory requirements, by local regulations, or by an agreement with Gilead. The investigator must notify Gilead before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead must be notified in advance.

If the investigator cannot provide for this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead to store these records securely away from the site so that they can be returned sealed to the investigator in case of an inspection. When source documents are required for the continued care of the subject, appropriate copies should be made for storage away from the site.

# 9.1.6. Case Report Forms

For each subject consented, an eCRF will be completed by an authorized study staff member whose training for this function is documented according to study procedures. eCRF should be completed on the day of the subject visit to enable the sponsor to perform central monitoring of safety data. Subsequent to data entry, a study monitor will perform source data verification within the EDC system. Original entries as well as any changes to data fields will be stored in the audit trail of the system. Prior to database lock (or any interim time points as described in the clinical data management plan), the investigator will used his/her log in credentials to confirm that the forms have been reviewed, and that the entries required per the protocol scheduled of events and procedures. System-generated or manual queries will be issued to the investigative site staff as data discrepancies are identified by the monitor or internal Gilead staff, who routinely review the data for completeness, correctness, and consistency. The site coordinator is responsible for responding to the queries in a timely manner, within the system, either by confirming the data as correct or updating the original entry, and providing the reason for the update (e.g. data entry error). At the conclusion of the trial, Gilead will provide the site with a read-only archive copy of the data entered by that site. This archive must be stored in accordance with the records retention requirements outlined in Section 9.1.5.

### 9.1.7. Investigational Medicinal Product Accountability and Return

Gilead recommends that used and unused IMP supplies be returned to the shipping facility from which it came for eventual destruction. The study monitor will provide instructions for return. If return is not possible, the study monitor will evaluate each study center's IMP disposal procedures and provide appropriate instruction for destruction of unused IMP supplies. If the site has an appropriate standard operating procedure (SOP) for drug destruction as determined by Gilead (Quality Assurance) QA, the site may destroy used (empty or partially empty) and unused IMP supplies in accordance with that site's approved SOP. A copy of the site's approved SOP will be obtained for central files.

If IMP is destroyed on site, the investigator must maintain accurate records for all IMP destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and the person who disposed of the IMP. Upon study completion, copies of the IMP accountability records must be filed at the site. Another copy will be returned to Gilead.

The study monitor will review IMP supplies and associated records at periodic intervals.

#### 9.1.8. Inspections

The investigator will make available all source documents and other records for this trial to Gilead's appointed study monitors, to IRBs [or] IECs, or to regulatory authority or health authority inspectors.

## 9.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

# 9.2. Sponsor Responsibilities

#### 9.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead. The investigator must submit all protocol modifications to the IRB [or] IEC in accordance with local requirements and receive documented IRB [or] IEC approval before modifications can be implemented.

#### 9.2.2. Study Report and Publications

A clinical study report (CSR) will be prepared and provided to the regulatory agencies. Gilead will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

- The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form or the study has been completed at all study sites for at least 2 years
- The investigator will submit to Gilead any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation.
- No such communication, presentation, or publication will include Gilead's confidential information (see Section 9.1.4).
- The investigator will comply with Gilead's request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

#### 9.3. Joint Investigator/Sponsor Responsibilities

#### 9.3.1. Access to Information for Monitoring

In accordance with regulations and guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the accuracy of the data recorded in the CRF/eCRF.

The monitor is responsible for routine review of the CRF/eCRF at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to verify the entries on the CRF/eCRF. The investigator agrees to cooperate with the monitor to ensure that any problems detected through any type of monitoring (central, on site) are resolved.

## 9.3.2. Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify the Gilead medical monitor immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead access to records, facilities, and personnel for the effective conduct of any inspection or audit.

## 9.3.3. Study Discontinuation

Both the sponsor and the investigator reserve the right to terminate the study at any time. Should this be necessary, both parties will arrange discontinuation procedures and notify the appropriate regulatory authority(ies), IRBs, and IECs. In terminating the study, Gilead and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.
# 10. REFERENCES

- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.
- Falck-Ytter Y, Kale H, Mullen KD, Sarbah SA, Sorescu L, McCullough AJ. Surprisingly small effect of antiviral treatment in patients with hepatitis C. Ann Intern Med 2002;136 (4):288-92.
- Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med 2001;345 (1):41-52.
- Yu JW, Wang GQ, Sun LJ, Li XG, Li SC. Predictive value of rapid virological response and early virological response on sustained virological response in HCV patients treated with pegylated interferon alpha-2a and ribavirin. J Gastroenterol Hepatol 2007;22 (6):832-6.
- Roche Pharmaceuticals. PEGASYS® (peginterferon alfa-2a). US Prescribing Information. Nutley, NJ. March 2010:
- Poordad F, McCone J, Jr., Bacon BR, Bruno S, Manns MP, Sulkowski MS, et al. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med 2011;364 (13):1195-206.
- Muir AJ, Provenzale D. A descriptive evaluation of eligibility for therapy among veterans with chronic hepatitis C virus infection. J Clin Gastroenterol 2002;34 (3):268-71.
- Backus LI, Boothroyd DB, Phillips BR, Mole LA. Predictors of response of US veterans to treatment for the hepatitis C virus. Hepatology 2007;46 (1):37-47.
- Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, et al. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med 2011;364 (25):2405-16.
- Sievert W, Altraif I, Razavi HA, Abdo A, Ahmed EA, Alomair A, et al. A systematic review of hepatitis C virus epidemiology in Asia, Australia and Egypt. Liver Int 2011;31 Suppl 2:61-80.
- Alter HJ, Liang TJ. Hepatitis C: the end of the beginning and possibly the beginning of the end. Ann Intern Med 2012;156 (4):317-8.
- 20839 Clopper CJ, Pearson ES. The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Dec. Biometrika 1934;26 (4):pp. 404-13.

- Al-Batran SE, Pauligk C, Wirtz R, Werner D, Steinmetz K, Homann N, et al. The validation of matrix metalloproteinase-9 mRNA gene expression as a predictor of outcome in patients with metastatic gastric cancer. Ann Oncol 2012;23 (7):1699-705.
- Ge D, Fellay J, Thompson AJ, Simon JS, Shianna KV, Urban TJ, et al. Genetic variation in IL28B predicts hepatitis C treatment-induced viral clearance. Nature 2009;461 (7262):399-401.
- Ghany MG, Strader DB, Thomas DL, Seeff LB. DO NOT USE Diagnosis, management, and treatment of hepatitis C: an update. Hepatology 2009;49 (4):1335-74.
- Nakano T, Lau GM, Sugiyama M, Mizokami M. An updated analysis of hepatitis C virus genotypes and subtypes based on the complete coding region. Liver Int 2012;32 (2):339-45.
- Thomas DL, Thio CL, Martin MP, Qi Y, Ge D, O'Huigin C, et al. Genetic variation in IL28B and spontaneous clearance of hepatitis C virus. Nature 2009;461 (7265):798-801.
- Thein HH, Yi Q, Dore GJ, Krahn MD. Estimation of stage-specific fibrosis progression rates in chronic hepatitis C virus infection: a meta-analysis and meta-regression. Hepatology 2008;48 (2):418-31.
- Tanaka Y, Nishida N, Sugiyama M, Kurosaki M, Matsuura K, Sakamoto N, et al. Genome-wide association of IL28B with response to pegylated interferon-alpha and ribavirin therapy for chronic hepatitis C. Nature genetics 2009;41 (10):1105-9.
- Negro F, Alberti A. The global health burden of hepatitis C virus infection. Liver Int 2011;31 Suppl 2:1-3.
- Omata M, Kanda T, Yu ML, Yokosuka O, Lim SG, al e. APASL consensus statements and management algorithms for hepatitis C virus infection. Hepatol International 2012;6:409-35.
- Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL, Jr., et al. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med 2002;347 (13):975-82.
- Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, et al. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet 2001;358 (9286):958-65.
- Huh K, Choi SY, Whang YS, Lee DS. Prevalence of viral hepatitis markers in Korean patients with hepatocellular carcinoma. J Korean Med Sci 1998;13 (3):306-10.

- 24209 Kim YS, Ahn YO, Lee HS. Risk factors for hepatitis C virus infection among Koreans according to the hepatitis C virus genotype. J Korean Med Sci 2002;17 (2):187-92.
- Lee HS, Han CJ, Kim CY. Predominant etiologic association of hepatitis C virus with hepatocellular carcinoma compared with hepatitis B virus in elderly patients in a hepatitis B-endemic area. Cancer 1993;72 (9):2564-7.
- Lim YS. Current status of liver disease in Korea: hepatitis C. The Korean journal of hepatology 2009;15 Suppl 6:S25-8.
- Lyoo K, Song MJ, Hur W, Choi JE, Hong SW, Kim CW, et al. Polymorphism near the IL28B gene in Korean hepatitis C virus-infected patients treated with peg-interferon plus ribavirin. J Clin Virol 2011;52 (4):363-6.
- Shin HR, Kim JY, Kim JI, Lee DH, Yoo KY, Lee DS, et al. Hepatitis B and C virus prevalence in a rural area of South Korea: the role of acupuncture. Br J Cancer 2002;87 (3):314-8.
- Shin HR. Epidemiology of hepatitis C virus in Korea. Intervirology 2006;49 (1-2):18-22.
- Suh DJ, Jeong SH. Current status of hepatitis C virus infection in Korea. Intervirology 2006;49 (1-2):70-5.
- Wei L, Lopez-Talavera JC, Rao H, Shang J, Chen H, Li J, et al. Prevalence of HCV Viral and Host IL28B Genotypes in China [Poster 412]. The Liver Meeting 2011: The 623nd Annual Meeting of the American Association for the Study of LIver Diseases; 2011 November 4-8; San Francisco, CA. Bristol-Myers Squibb.
- Yu ML, Chuang WL. Treatment of chronic hepatitis C in Asia: when East meets West. J Gastroenterol Hepatol 2009;24 (3):336-45.
- 24235 Chen CH, Yang PM, Huang GT, Lee HS, Sung JL, Sheu JC. Estimation of seroprevalence of hepatitis B virus and hepatitis C virus in Taiwan from a large-scale survey of free hepatitis screening participants. J Formos Med Assoc 2007;106 (2):148-55.
- Heo N-Y, Lim Y-S, Lee HC, Lee YS, Kim KM, Byum KS, et al. High effectiveness of peginterferon alfa-2a plus ribavirin therapy in Korean patients with chronic hepatitis C in clinical practice. Clin Mol Hepatol 2013;19 (1):60-9.
- Lee H, Choi MS, Paik SW, Kim JH, Kim DY, Lee JH, et al. [Peginterferon alfa-2a plus ribavirin for initial treatment of chronic hepatitis C in Korea]. The Korean journal of hepatology 2006;12 (1):31-40.
- 24238 Sinn DH, Kim YJ, Lee ST, Gwak GY, Choi MS, Lee JH, et al. Association of a single nucleotide polymorphism near the interleukin-28B gene with response to hepatitis C therapy in Asian patients. J Gastroenterol Hepatol 2011;26 (9):1374-9.

- Huang JF, Yu ML, Huang CF, Chiu CF, Dai CY, Huang CI, et al. The efficacy and safety of pegylated interferon plus ribavirin combination therapy in chronic hepatitis c patients with hepatocellular carcinoma post curative therapies a multicenter prospective trial. J Hepatol 2011;54 (2):219-26.
- Lin CY, Chen JY, Lin TN, Jeng WJ, Huang CH, Huang CW, et al. IL28B SNP rs12979860 is a critical predictor for on-treatment and sustained virologic response in patients with hepatitis C virus genotype-1 infection. PLoS ONE 2011;6 (3):e18322.
- Yu ML, Huang CF, Huang JF, Chang NC, Yang JF, Lin ZY, et al. Role of interleukin-28B polymorphisms in the treatment of hepatitis C virus genotype 2 infection in Asian patients. Hepatology 2011;53 (1):7-13.
- Liu CH, Liu CJ, Lin CL, Liang CC, Hsu SJ, Yang SS, et al. Pegylated interferonalpha-2a plus ribavirin for treatment-naive Asian patients with hepatitis C virus genotype 1 infection: a multicenter, randomized controlled trial. Clin Infect Dis 2008;47 (10):1260-9.
- Lee HJ, Eun JR, Choi JW, Kim KO, Moon HJ. [Comparison of therapeutic results between combination therapy of peginterferon alpha-2a plus ribavirin and interferon alpha-2b plus ribavirin according to treatment duration in patients with chronic hepatitis C]. The Korean journal of hepatology 2008;14 (1):46-57.
- Kim JI, Kim SH, Lee BS, Lee HY, Lee TH, Kang YW, et al. [Efficacy of initial treatment with peginterferon alpha-2a versus peginterferon alpha-2b in combination with ribavirin in naive chronic hepatitis C patients living in Daejeon and Chungcheong Province in Korea: a comparative study]. The Korean journal of hepatology 2008;14 (4):493-502.
- Jun DW, Tak WY, Bae SH, Lee YJ. Recent trends in the treatment of chronic hepatitis C. The Korean journal of hepatology 2012;18 (1):22-8.
- Huang CF, Yang JF, Dai CY, Huang JF, Hou NJ, Hsieh MY, et al. Efficacy and safety of pegylated interferon combined with ribavirin for the treatment of older patients with chronic hepatitis C. J Infect Dis 2010;201 (5):751-9.
- Guo X, Zhao Z, Xie J, Cai Q, Zhang X, Peng L, et al. Prediction of response to pegylated-interferon-alpha and ribavirin therapy in Chinese patients infected with different hepatitis C virus genotype. Virology journal 2012;9:123.
- Gao X, Cui Q, Shi X, Su J, Peng Z, Chen X, et al. Prevalence and trend of hepatitis C virus infection among blood donors in Chinese mainland: a systematic review and meta-analysis. BMC Infect Dis 2011;11:88.
- Marcus EL, Tur-Kaspa R. Chronic hepatitis C virus infection in older adults. Clin Infect Dis 2005;41 (11):1606-12.

- Kim KT, Han SY, Kim JH, Yoon HA, Baek YH, Kim MJ, et al. [Clinical outcome of pegylated interferon and ribavirin therapy for chronic hepatitis C]. The Korean journal of hepatology 2008;14 (1):36-45.
- Cheong HR, Woo HY, Heo J, Yoon KT, Kim DU, Kim GH, et al. [Clinical efficacy and safety of the combination therapy of peginterferon alpha and ribavirin in cirrhotic patients with HCV infection]. The Korean journal of hepatology 2010;16 (1):38-48.
- Zheng YY, Fan XH, Wang LF, Tian D, Huo N, Lu HY, et al. Efficacy of pegylated interferon-alpha-2a plus ribavirin for patients aged at least 60 years with chronic hepatitis C. Chinese medical journal 2012;125 (11):1852-6.
- Yu ML, Dai CY, Lin ZY, Lee LP, Hou NJ, Hsieh MY, et al. A randomized trial of 24- vs. 48-week courses of PEG interferon alpha-2b plus ribavirin for genotype-1b-infected chronic hepatitis C patients: a pilot study in Taiwan. Liver Int 2006;26 (1):73-81.
- The Chinese Society of Hepatology of the Chinese Medical Association.
  Guidelines for Hepatitis C Prevention and Treatment. Chin J Prev Med 2004;38
  (3).
- Kang MJ, Jung EU, Park SW, Choi P, Kim JH, Park SJ, et al. [Effects of pegylated interferon and ribavirin in Korean patients with chronic hepatitis C virus infection]. The Korean journal of hepatology 2008;14 (3):318-30.
- McCaughan GW, Omata M, Amarapurkar D, Bowden S, Chow WC, Chutaputti A, et al. Asian Pacific Association for the Study of the Liver consensus statements on the diagnosis, management and treatment of hepatitis C virus infection. J Gastroenterol Hepatol 2007;22 (5):615-33.
- Zhou BT, Fan YM, Li TM, Liu XQ. [Effectiveness of combined therapies using two types of peginterferon and ribavirin in treating chronic hepatitis C virus genotypes 1b/6a infections]. Zhongguo yi xue ke xue yuan xue bao. Acta Academiae Medicinae Sinicae 2010;32 (3):320-3.
- 25091 Schaefer M, Mauss S. Hepatitis C treatment in patients with drug addiction: clinical management of interferon-alpha-associated psychiatric side effects. Current drug abuse reviews 2008;1 (2):177-87.
- Shang G, Seed CR, Wang F, Nie D, Farrugia A. Residual risk of transfusion-transmitted viral infections in Shenzhen, China, 2001 through 2004. Transfusion 2007;47 (3):529-39.
- Zhou Y, Wang X, Mao Q, Fan Y, Zhu Y, Zhang X, et al. Changes in modes of hepatitis C infection acquisition and genotypes in southwest China. J Clin Virol 2009;46 (3):230-3.

- 25095 Huang C, Qiu F, Guo M, Yi Y, Shen L, Wang F, et al. Prevalence and risk factors of hepatitis C among former blood donors in rural China. Int J Infect Dis 2012;16 (10):e731-4.
- Weir MR. Renal effects of nonselective NSAIDs and coxibs. Cleve Clin J Med 2002;69 Suppl 1:SI53-8.
- Yilmaz A, Price RW, Gisslen M. Antiretroviral drug treatment of CNS HIV-1 infection. J Antimicrob Chemother 2012;67 (2):299-311.
- Jin YJ, Lee JW, Lee JI, Park SH, Park CK, Kim YS, et al. Multicenter comparison of PEG-IFN alpha2a or alpha2b plus ribavirin for treatment-naive HCV patient in Korean population. BMC gastroenterology 2013;13:74.
- Kim HI, Kim IH, Jeon BJ, Lee S, Kim SH, Kim SW, et al. Treatment Response and Tolerability of Pegylated Interferon-alpha Plus Ribavirin Combination Therapy in elderly Patients (>/= 65 years) With Chronic Hepatitis C in Korea. Hepat Mon 2012;12 (7):430-6.
- Park SY, Rim MY, Yo IK, Ha MS, Kim JS, Lee JW, et al. [Efficacy of peginterferon and ribavirin combination therapy of chronic hepatitis C: a pooled analysis]. The Korean journal of gastroenterology = Taehan Sohwagi Hakhoe chi 2012;60 (5):306-14.
- Sun CA, Chen HC, Lu CF, You SL, Mau YC, Ho MS, et al. Transmission of hepatitis C virus in Taiwan: prevalence and risk factors based on a nationwide survey. J Med Virol 1999;59 (3):290-6.
- Yu ML, Chuang WL, Chen SC, Dai CY, Hou C, Wang JH, et al. Changing prevalence of hepatitis C virus genotypes: molecular epidemiology and clinical implications in the hepatitis C virus hyperendemic areas and a tertiary referral center in Taiwan. J Med Virol 2001;65 (1):58-65.
- 29247 Lee CM, Lu SN, Hung CH, Tung WC, Wang JH, Tung HD, et al. Hepatitis C virus genotypes in southern Taiwan: prevalence and clinical implications. Trans R Soc Trop Med Hyg 2006;100 (8):767-74.
- Sun CA, Chen HC, Lu SN, Chen CJ, Lu CF, You SL, et al. Persistent hyperendemicity of hepatitis C virus infection in Taiwan: the important role of iatrogenic risk factors. J Med Virol 2001;65 (1):30-4.

# 11. APPENDICES

| Appendix 1. | Investigator Signature Page |
|---|---|
| Appendix 2. | Study Procedures Table |
| Appendix 3. | GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities |
| Appendix 4. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and |
| | Contraceptive Requirements |
| Appendix 5. | Calculation of Historical Control SVR12 for Treatment-naïve Korean Subjects and |
| | for Treatment-naïve Chinese Subjects with Chronic GT-1 HCV Infection |

## Appendix 1.

**Investigator Signature Page** 

# GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE FOSTER CITY, CA 94404

#### STUDY ACKNOWLEDGEMENT

A Phase 3b, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination in Treatment-Naïve and Treatment-Experienced Subjects with Chronic Genotype 1 HCV Infection

# GS-US-337-0131, Amendment 3.0, 12 February 2016

| GS-US-337-0131, Amendment 3.0, 12 February 2016 | |
|---|---|
| This protocol has been approved by Gilead Sciences, Inc. The following signature document this approval. | ts |
| Jenny Yang/PharmD (Printed) Study Director | |
| Date INVESTIGATOR STATEMENT | |

I have read the protocol, including all appendices, and I agree that it contains all necessary details for me and my staff to conduct this study as described. I will conduct this study as outlined herein and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and access to all information provided by Gilead Sciences, Inc. I will discuss this material with them to ensure that they are fully informed about the drugs and the study.

| Principal Investigator Name (Printed) | Signature | |
|---------------------------------------|-------------|--------|
| Date | Site Number | No. of |

# **Appendix 2. Study Procedures Table**

# Table 1. Screening and On-Treatment Study Visits

| | On Treatment Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Clinical Assessments | Day -28<br>to Day -1 | Baseline/<br>Day 1 <sup>b</sup> | Week 1<br>(±3 days) | Week 2<br>(±3 days) | Week 4<br>(±3 days) | Week 6<br>(±3 days) | Week 8<br>(±3 days) | Week 10<br>(±3 days) | Week 12<br>(±3 days) | ET |
| Informed Consent | X | | | | | | | | | |
| Determine Eligibility | X | X | | | | | | | | |
| Medical History | X | | | | | | | | | |
| Physical Examination | X | X | | | | | | | X | X |
| Liver Imaging (Cirrhotics Only) | X | | | | | | | | | |
| Height | X | | | | | | | | | |
| Weight | X | X | | | | | | | X | X |
| Vital Signs <sup>c</sup> | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>d</sup> | X | X | X | | | | | | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Prevention<br>Counseling | | X | | | | | | | X | X |
| Health Related Quality of Life | | X | | X | X | | X | | X | X |
| Hematology & Chemistry | X | X | X | X | X | X | X | X | X | X |
| Coagulation | X | X | | | | | | | X | X |
| Serum HCV RNA | X | X | X | X | X | X | X | X | X | X |

| | On Treatment Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Clinical Assessments | Day -28<br>to Day -1 | Baseline/<br>Day 1 <sup>b</sup> | Week 1<br>(±3 days) | Week 2<br>(±3 days) | Week 4<br>(±3 days) | Week 6<br>(±3 days) | Week 8<br>(±3 days) | Week 10<br>(±3 days) | Week 12<br>(±3 days) | ET |
| Single PK Sample | | | X | X | X | X | X | X | X | X |
| Viral RNA Sequencing /Phenotyping Sample (Plasma) <sup>e</sup> | | X | X | X | X | X | X | X | X | X |
| Archive Sample <sup>j</sup> | | X | | | | | | | X | X |
| Serum or Urine Pregnancy Test <sup>k</sup> | X | X | | | X | | X | | X | X |
| Urinalysis | X | | | | | | | | | |
| IL28B Genotype, HCV<br>Genotype | X | | | | | | | | | |
| HCV Ab, HIV Ab and HBsAg | X | | | | | | | | | |
| Hemoglobin A1c, TSH | X | | | | | | | | | |
| PK Substudy Collection <sup>f</sup> | | | | X | X | | | | | |
| Single Pharmacogenomic Sample <sup>g</sup> | | X | | | | | | | | |
| Review of Study Drug<br>Adherence and Drug<br>Accountability <sup>h</sup> | | | X | X | X | X | X | X | X | X |
| Study Drug Dispensing <sup>i</sup> | | X | | | X | | X | | | |

a The screening window can be extended to 42 days for subjects requiring liver biopsy or additional HCV genotype testing.

b Baseline/Day 1 assessments must be performed prior to dosing.

c Vital signs include resting blood pressure, pulse, respiratory rate and temperature.

d Subjects will be required to rest in a supine position for  $\geq 5$  minutes prior to making a recording. The investigator (or qualified designee) should review the ECG traces recorded in real time for gross abnormalities.

e Serum samples will be collected and stored for potential HCV sequencing and other virology studies.

- f The optional PK substudy is conducted in Taiwan and Korea only. Subjects that consent to the optional PK substudy will have serial PK samples drawn at Week 2 or Week 4 visit.
- g Only for subjects who have provided consent for this sample and testing (Taiwan and Korea only). This sample can be obtained at a subsequent visit if not obtained at Day 1.
- h Study medication and dosing diary, will be reconciled at every post-baseline visit by the investigator or designee in order to monitor the subject's adherence with the medication regimen.
- i Study Drug will be dispensed per IWRS directions. Subjects must be instructed to bring back all bottles of study medication(s) in the original container at every post baseline study visits through the end of treatment.
- j Archive plasma samples will be collected at the Baseline/Day 1 visit and at the end of treatment for subjects who have not opted out of sample collection.
- k For female subjects of childbearing potential. In the event of a positive urine test, a serum pregnancy test will be done.

Table 2. Post Treatment Study Visits

| | | Post Treatment Period <sup>a</sup> | |
|---|---|---|---|
| Clinical Assessments | Post Treatment Week 4<br>(±5 days) | Post Treatment Week 12<br>(±5 days) | Post Treatment Week 24<br>(±5 days) |
| Weight | | X | X |
| Vital Signs <sup>b</sup> | X | X | X |
| Adverse Events | X | | |
| Concomitant Medications | X | | |
| Pregnancy Prevention Counseling | X | | |
| Health Related Quality of Life | X | X | |
| Hematology & Chemistry | X | | |
| Serum HCV RNA | X | X | X |
| Viral Sequencing Sample (Plasma) <sup>c</sup> | X | X | X |
| Serum or Urine Pregnancy Test <sup>d</sup> | X | | |

a All subjects will complete both 4-week and 12-week Post-Treatment visits regardless of the treatment duration. Subjects with HCV RNA < LLOQ at their 12-week Post-Treatment visit will complete a 24-week Post-Treatment visit, unless viral relapse is determined. The end of study will occur at the 24-week Post-Treatment visit.

b Vital signs include resting blood pressure, pulse, respiratory rate and temperature.

c Plasma samples will be collected and stored for potential HCV sequencing and other virology studies.

d For female subjects of childbearing potential. In the event of a positive urine test, a serum pregnancy test will be done.

Appendix 3. GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities

Version: 18June2012

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin<br>HIV POSITIVE | 8.5 to 10.0 g/dL | 7.5 to < 8.5 g/dL | 6.5 to < 7.5 g/dL | < 6.5 g/dL |
| Adult and Pediatric ≥ 57 Days | 85 to 100 g/L | 75 to < 85 g/L | 65 to < 75 g/L | < 65 g/L |
| HIV NEGATIVE | 10.0 to 10.9 g/dL | 9.0 to < 10.0 g/dL | 7.0 to < 9.0 g/dL | < 7.0 g/dL |
| Adult and Pediatric ≥ 57 Days | 100 to 109 g/L | 90 to < 100 g/L | 70 to < 90 g/L | < 70 g/L |
| | OR | OR | OR | |
| | Any decrease from Baseline | Any decrease from Baseline | Any decrease from Baseline | |
| | 2.5 to < 3.5 g/dL | 3.5 to < 4.5 g/dL | ≥ 4.5 g/dL | |
| | 25 to < 35 g/L | 35 to < 45 g/L | ≥ 45 g/L | |
| Infant, 36–56 Days | 8.5 to 9.4 g/dL | 7.0 to < 8.5 g/dL | 6.0 to < 7.0 g/dL | < 6.0 g/dL |
| (HIV <u>POSITIVE</u> OR <u>NEGATIVE</u> ) | 85 to 94 g/L | 70 to < 85 g/L | 60 to < 70 g/L | < 60 g/L |
| Infant, 22–35 Days | 9.5 to 10.5 g/dL | 8.0 to < 9.5 g/dL | 7.0 to < 8.0 g/dL | < 7.0 g/dL |
| (HIV <u>POSITIVE</u> OR <u>NEGATIVE</u> ) | 95 to 105 g/L | 80 to < 95 g/L | 70 to < 80 g/L | < 70 g/L |
| Infant, 1–21 Days | 12.0 to 13.0 g/dL | 10.0 to < 12.0 g/dL | 9.0 to < 10.0 g/dL | < 9.0 g/dL |
| (HIV <u>POSITIVE</u> OR <u>NEGATIVE</u> ) | 120 to 130 g/L | 100 to < 120 g/L | 90 to < 100 g/L | < 90 g/L |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Absolute Neutrophil Count (ANC) | 1000 to 1300/mm <sup>3</sup> | 750 to < 1000/mm <sup>3</sup> | 500 to < 750/mm <sup>3</sup> | < 500/mm <sup>3</sup> |
| Adult and Pediatric, > 7 Days | 1.00 to 1.30 GI/L | 0.75 to < 1.00 GI/L | 0.50 to < 0.75 GI/L | < 0.50 GI/L |
| Infant, 2 – ≤ 7 Days | 1250 to 1500/mm <sup>3</sup> | 1000 to < 1250/mm <sup>3</sup> | 750 to < 1000/mm <sup>3</sup> | < 750/mm <sup>3</sup> |
| | 1.25 to 1.50 GI/L | 1.00 to < 1.25 GI/L | 0.75 to < 1.00 GI/L | < 0.75 GI/L |
| Infant, 1 Day | 4000 to 5000/mm <sup>3</sup> | 3000 to < 4000/mm <sup>3</sup> | 1500 to < 3000/mm <sup>3</sup> | < 1500/mm <sup>3</sup> |
| | 4.00 to 5.00 GI/L | 3.00 to < 4.00 GI/L | 1.50 to < 3.00 GI/L | < 1.50 GI/L |
| Absolute CD4+ Count | | | | |
| HIV NEGATIVE ONLY | | | | |
| Adult and Pediatric | 300 to 400/mm <sup>3</sup> | 200 to < 300/mm <sup>3</sup> | $100 \text{ to} < 200/\text{mm}^3$ | < 100/mm <sup>3</sup> |
| > 13 Years | 300 to 400/μL | $200 \text{ to} < 300/\mu\text{L}$ | $100 \text{ to} < 200/\mu\text{L}$ | < 100/μL |
| Absolute Lymphocyte Count | | | | |
| HIV NEGATIVE ONLY | | | | |
| Adult and Pediatric | 600 to 650/mm <sup>3</sup> | 500 to < 600/mm <sup>3</sup> | 350 to < 500/mm <sup>3</sup> | < 350/mm <sup>3</sup> |
| > 13 Years | 0.60 to 0.65 GI/L | 0.50 to < 0.60 GI/L | 0.35 to < 0.50 GI/L | < 0.35 GI/L |
| Platelets | 100,000 to < 125,000/mm <sup>3</sup> | 50,000 to < 100,000/mm <sup>3</sup> | 25,000 to < 50,000/mm <sup>3</sup> | < 25,000/mm <sup>3</sup> |
| | 100 to < 125 GI/L | 50 to < 100 GI/L | 25 to < 50 GI/L | < 25 GI/L |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| WBCs | 2000/mm <sup>3</sup> to 2500/mm <sup>3</sup> | 1,500 to < 2,000/mm <sup>3</sup> | 1000 to < 1,500/mm <sup>3</sup> | < 1000/mm <sup>3</sup> |
| | 2.00 GI/L to 2.50 GI/L | 1.50 to < 2.00 GI/L | 1.00 to < 1.50 GI/L | < 1.00 GI/L |
| Hypofibrinogenemia | 100 to 200 mg/dL | 75 to < 100 mg/dL | 50 to < 75 mg/dL | < 50 mg/dL |
| | 1.00 to 2.00 g/L | 0.75 to < 1.00 g/L | 0.50 to < 0.75 g/L | < 0.50 g/L |
| Hyperfibrinogenemia | > ULN to 600 mg/dL | > 600 mg/dL | _ | _ |
| | > ULN to 6.0 g/L | > 6.0 g/L | _ | _ |
| Fibrin Split Product | 20 to 40 μg/mL | > 40 to 50 μg/mL | > 50 to 60 μg/mL | > 60 μg/mL |
| | 20 to 40 mg/L | > 40 to 50 mg/L | > 50 to 60 mg/L | > 60 mg/L |
| Prothrombin Time (PT) | > 1.00 to 1.25 × ULN | > 1.25 to 1.50 × ULN | > 1.50 to 3.00 × ULN | > 3.00 × ULN |
| International Normalized Ratio of prothrombin time (INR) | 1.1 to 1.5 x ULN | >1.5 to 2.0 x ULN | >2.0 to 3.0 x ULN | >3.0 x ULN |
| Activated Partial | | | | |
| Thromboplastin Time (APTT) | > 1.00 to 1.66 × ULN | > 1.66 to 2.33 × ULN | > 2.33 to 3.00 × ULN | > 3.00 × ULN |
| Methemoglobin | 5.0 to 10.0% | > 10.0 to 15.0% | > 15.0 to 20.0% | > 20.0% |

| | CHEMISTRY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to <lln l<="" meq="" td=""><td>125 to &lt; 130 mEq/L</td><td>121 to &lt; 125 mEq/L</td><td>&lt; 121 mEq/L</td></lln> | 125 to < 130 mEq/L | 121 to < 125 mEq/L | < 121 mEq/L |
| | 130 to <lln l<="" mmol="" td=""><td>125 to &lt; 130 mmol/L</td><td>121 to &lt; 125 mmol/L</td><td>&lt; 121 mmol/L</td></lln> | 125 to < 130 mmol/L | 121 to < 125 mmol/L | < 121 mmol/L |
| Hypernatremia | 146 to 150 mEq/L | > 150 to 154 mEq/L | > 154 to 159 mEq/L | > 159 mEq/L |
| | 146 to 150 mmol/L | > 150 to 154 mmol/L | > 154 to 159 mmol/L | > 159 mmol/L |
| Hypokalemia | 3.0 to 3.4 mEq/L | 2.5 to < 3.0 mEq/L | 2.0 to < 2.5 mEq/L | < 2.0 mEq/L |
| | 3.0 to 3.4 mmol/L | 2.5 to < 3.0 mmol/L | 2.0 to < 2.5 mmol/L | < 2.0 mmol/L |
| Hyperkalemia | 5.6 to 6.0 mEq/L | > 6.0 to 6.5 mEq/L | > 6.5 to 7.0 mEq/L | > 7.0 mEq/L |
| | 5.6 to 6.0 mmol/L | > 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mmol/L | > 7.0 mmol/L |
| Hypoglycemia | | | | |
| Adult and Pediatric | 55 to 64 mg/dL | 40 to < 55 mg/dL | 30 to < 40 mg/dL | < 30 mg/dL |
| | 3.03 to 3.58 mmol/L | 2.20 to < 3.03 mmol/L | 1.64 to < 2.20 mmol/L | < 1.64 mmol/L |
| ≥ 1 Month<br>Infant,< 1 Month | 50 to 54 mg/dL | 40 to < 50 mg/dL | 30 to < 40 mg/dL | < 30 mg/dL |
| | 2.8 to 3.0 mmol/L | 2.2 to < 2.8 mmol/L | 1.7 to < 2.2 mmol/L | < 1.7 mmol/L |
| Hyperglycemia, Nonfasting | 116 to 160 mg/dL | > 160 to 250 mg/dL | > 250 to 500 mg/dL | > 500 mg/dL |
| | 6.42 to 8.91 mmol/L | > 8.91 to 13.90 mmol/L | > 13.90 to 27.79 mmol/L | > 27.79 mmol/L |
| Hyperglycemia, Fasting | 110 to 125 mg/dL | >125 to 250 mg/dL | >250 to 500 mg/dL | >500 mg/dL |
| | 6.08 to 6.96 mmol/L | >6.96 to 13.90 mmol/L | >13.90 to 27.79 mmol/L | >27.79 mmol/L |

| | CHEMISTRY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypocalcemia | | | | |
| (corrected for albumin if appropriate*) | 7.8 to 8.4 mg/dL<br>1.94 to 2.10 mmol/L | 7.0 to < 7.8 mg/dL<br>1.74 to < 1.94 mmol/L | 6.1 to < 7.0 mg/dL<br>1.51 to < 1.74 mmol/L | < 6.1 mg/dL<br>< 1.51 mmol/L |
| Adult and Pediatric | | | | |
| ≥7 Days<br>Infant, <7 Days | 6.5 to 7.5 mg/dL | 6.0 to < 6.5 mg/dL | 5.5 to < 6.0 mg/dL | < 5.5 mg/dL |
| | 1.61 to 1.88 mmol/L | 1.49 to < 1.61 mmol/L | 1.36 to < 1.49 mmol/L | < 1.36 mmol/L |
| Hypercalcemia (corrected for albumin if appropriate*) Adult and Pediatric ≥ 7 Days | >ULN to 11.5 mg/dL<br>>ULN to 2.88 mmol/L | > 11.5 to 12.5 mg/dL<br>> 2.88 to 3.13 mmol/L | > 12.5 to 13.5 mg/dL<br>> 3.13 to 3.38 mmol/L | > 13.5 mg/dL<br>> 3.38 mmol/L |
| Infant, < 7 Days | 11.5 to 12.4 mg/dL 2.86 to 3.10 mmol/L | > 12.4 to 12.9 mg/dL<br>> 3.10 to 3.23 mmol/L | > 3.13 to 3.38 mmol/L<br>> 12.9 to 13.5 mg/dL<br>> 3.23 to 3.38 mmol/L | > 3.38 mmol/L<br>> 13.5 mg/dL<br>> 3.38 mmol/L |
| Hypocalcemia (ionized) | 3.0 mg/dL to < LLN<br>0.74 mmol/L to < LLN | 2.5 to < 3.0 mg/dL<br>0.62 to < 0.74 mmol/L | 2.0 to < 2.5 mg/dL<br>0.49 to < 0.62 mmol/L | < 2.0 mg/dL<br>< 0.49 mmol/L |
| Hypercalcemia (ionized) | > ULN to 6.0 mg/dL<br>> ULN to 1.50 mmol/L | > 6.0 to 6.5 mg/dL<br>> 1.50 to 1.63 mmol/L | > 6.5 to 7.0 mg/dL<br>> 1.63 to 1.75 mmol/L | > 7.0 mg/dL<br>> 1.75 mmol/L |

| | CHEMISTRY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypomagnesemia | 1.40 to <lln dl<="" mg="" td=""><td>1.04 to &lt; 1.40 mg/dL</td><td>0.67 to &lt; 1.04 mg/dL</td><td>&lt; 0.67 mg/dL</td></lln> | 1.04 to < 1.40 mg/dL | 0.67 to < 1.04 mg/dL | < 0.67 mg/dL |
| | 1.2 to <lln l<="" meq="" td=""><td>0.9 to &lt; 1.2 mEq/L</td><td>0.6 to &lt; 0.9 mEq/L</td><td>&lt; 0.6 mEq/L</td></lln> | 0.9 to < 1.2 mEq/L | 0.6 to < 0.9 mEq/L | < 0.6 mEq/L |
| | 0.58 to <lln l<="" mmol="" td=""><td>0.43 to &lt; 0.58 mmol/L</td><td>0.28 to &lt; 0.43 mmol/L</td><td>&lt; 0.28 mmol/L</td></lln> | 0.43 to < 0.58 mmol/L | 0.28 to < 0.43 mmol/L | < 0.28 mmol/L |
| Hypophosphatemia | | | | |
| Adult and Pediatric | 2.0 to < LLN mg/dL | 1.5 to < 2.0 mg/dL | 1.0 to < 1.5 mg/dL | < 1.0 mg/dL |
| > 14 Years | 0.63 to < LLN mmol/L | 0.47 to < 0.63 mmol/L | 0.31 to < 0.47 mmol/L | < 0.31 mmol/L |
| Pediatric 1 Year–14 Years | 3.0 to 3.5 mg/dL | 2.5 to < 3.0 mg/dL | 1.5 to < 2.5 mg/dL | < 1.5 mg/dL |
| | 0.96 to 1.14 mmol/L | 0.80 to < 0.96 mmol/L | 0.47 to < 0.80 mmol/L | < 0.47 mmol/L |
| Pediatric < 1 Year | 3.5 to 4.5 mg/dL | 2.5 to < 3.5 mg/dL | 1.5 to < 2.5 mg/dL | < 1.5 mg/dL |
| | 1.12 to 1.46 mmol/L | 0.80 to < 1.12 mmol/L | 0.47 to < 0.80 mmol/L | < 0.47 mmol/L |
| Hyperbilirubinemia | | | | |
| Adult and Pediatric > 14 Days | > 1.0 to 1.5 × ULN | > 1.5 to 2.5 × ULN | > 2.5 to 5.0 × ULN | > 5.0 × ULN |
| Infant, ≤ 14 Days (non-hemolytic) | NA | 20.0 to 25.0 mg/dL | > 25.0 to 30.0 mg/dL | > 30.0 mg/dL |
| (non-nemorytic) | | 342 to 428 μmol/L | > 428 to 513 μmol/L | > 513 μmol/L |
| Infant, ≤ 14 Days | NA | NA | 20.0 to 25.0 mg/dL | > 25.0 mg/dL |
| (hemolytic) | | | 342 to 428 μmol/L | > 428 μmol/L |
| Blood Urea Nitrogen | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Hyperuricemia | >ULN to 10.0 mg/dL | > 10.0 to 12.0 mg/dL | > 12.0 to 15.0 mg/dL | > 15.0 mg/dL |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| | >ULN to 597 μmol/L | > 597 to 716 μmol/L | > 716 to 895 μmol/L | > 895 μmol/L |
| Hypouricemia | 1.5 mg/dL to < LLN | 1.0 to < 1.5 mg/dL | 0.5 to < 1.0 mg/dL | < 0.5 mg/dL |
| | 87 μmol/L to < LLN | 57 to < 87 μmol/L | 27 to < 57 μmol/L | < 27 μmol/L |
| Creatinine | > 1.50 to 2.00 mg/dL | > 2.00 to 3.00 mg/dL | > 3.00 to 6.00 mg/dL | > 6.00 mg/dL |
| | > 133 to 177 μmol/L | > 177 to 265 μmol/L | > 265 to 530 μmol/L | > 530 μmol/L |
| Bicarbonate | 16.0 mEq/L to < LLN | 11.0 to < 16.0 mEq/L | 8.0 to < 11.0 mEq/L | < 8.0 mEq/L |
| | 16.0 mmol/L to < LLN | 11.0 to < 16.0 mmol/L | 8.0 to < 11.0 mmol/L | < 8.0 mmol/L |
| Triglycerides | NA | 500 to 750 mg/dL | > 750 to 1200 mg/dL | > 1200 mg/dL |
| (Fasting) | | 5.64–8.47 mmol/L | > 8.47–13.55 mmol/L | > 13.55 mmol/L |
| LDL | 130 to 160 mg/dL | >160 to 190 mg/dL | > 190 mg/dL | NA |
| (Fasting) | 3.35 to 4.15 mmol/L | >4.15 to 4.92 mmol/L | >4.92 mmol/L | |
| Pediatric >2 to <18 years | 110 to 130 mg/dL | >130 to 190 mg/dL | > 190 mg/dL | NA |
| | 2.84 to 3.37 mmol/L | >3.37 to 4.92 mmol/L | >4.92 mmol/L | |
| Hypercholesterolemia | 200 to 239 mg/dL | > 239 to 300 mg/dL | > 300 mg/dL | NA |
| (Fasting) | 5.16 to 6.19 mmol/L | > 6.19 to 7.77 mmol/L | > 7.77 mmol/L | |
| Pediatric < 18 Years | 170 to 199 mg/dL | > 199 to 300 mg/dL | > 300 mg/dL | NA |
| | 4.39 to 5.15 mmol/L | > 5.15 to 7.77 mmol/L | > 7.77 mmol/L | |
| Creatine Kinase | $3.0 \text{ to} < 6.0 \times \text{ULN}$ | 6.0 to < 10.0 × ULN | 10.0 to < 20.0 × ULN | ≥ 20.0 × ULN |

<sup>\*</sup> Calcium should be corrected for albumin if albumin is < 4.0 g/dL

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| ALT (SGPT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| GGT | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Alkaline Phosphatase | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Total Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Pancreatic Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Lipase | > 1.0 to 1.5 × ULN | > 1.5 to 3.0 × ULN | > 3.0 to 5.0 × ULN | > 5.0 × ULN |
| Albumin | 3.0 g/dL to < LLN | 2.0 to < 3.0 g/dL | < 2.0 g/dL | NA |
| | 30 g/L to < LLN | 20 to < 30 g/L | < 20 g/L | |

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hematuria (Dipstick) | 1+ | 2+ | 3-4+ | NA |
| Hematuria (Quantitative) | | | | |
| See Note below | | | | |
| Females | >ULN - 10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Males | 6-10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Proteinuria (Dipstick) | 1+ | 2–3+ | 4+ | NA |
| Proteinuria, 24 Hour Collection | | | | |
| Adult and Pediatric<br>≥ 10 Years | 200 to 999 mg/24 h | >999 to 1999 mg/24 h | >1999 to 3500 mg/24 h | > 3500 mg/24 h |
| Pediatric > 3 Mo to<br>< 10 Years | 201 to 499 mg/m <sup>2</sup> /24 h | >499 to 799 mg/m <sup>2</sup> /24 h | >799 to 1000 mg/m <sup>2</sup> /24 h | > 1000 mg/ m <sup>2</sup> /24 h |
| Glycosuria (Dipstick) | 1+ | 2-3+ | 4+ | NA |

#### Notes:

Toxicity grades for Quantitative and Dipstick Hematuria will be assigned by Covance Laboratory, however for other laboratories, toxicity grades will only be assigned to Dipstick Hematuria.

With the exception of lipid tests, any graded laboratory test with a result that is between the LLN and ULN should be assigned Grade 0.

If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE.

| | | CARDIOVASCULAR | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Arrhythmia (general) (By ECG or physical exam) | Asymptomatic AND No intervention indicated | Asymptomatic AND Non-<br>urgent medical intervention<br>indicated | Symptomatic, non-life-<br>threatening AND Non-<br>urgent medical intervention<br>indicated | Life-threatening arrhythmia<br>OR Urgent intervention<br>indicated |
| Cardiac-ischemia/Infarction | NA | NA | Symptomatic ischemia (stable angina) OR Testing consistent with ischemia | Unstable angina OR Acute myocardial infarction |
| Hemorrhage (significant acute blood loss) | NA | Symptomatic AND No transfusion indicated | Symptomatic AND Transfusion of ≤ 2 units packed RBCs (for children ≤ 10 cc/kg) indicated | Life-threatening hypotension<br>OR Transfusion of > 2 units<br>packed RBCs indicated (for<br>children ≤ 10 cc/kg) indicated |
| Hypertension (with repeat testing at same visit) | OR<br>90–99 mmHg diastolic | > 159–179 mmHg systolic<br>OR<br>> 99–109 mmHg diastolic | > 179 mmHg systolic<br>OR<br>> 109 mmHg diastolic | Life-threatening consequences (eg, malignant hypertension) OR Hospitalization (other than ER visit) indicated |
| Pediatric ≤ 17 Years (with repeat testing at same visit) | NA | 91st–94th percentile adjusted<br>for age, height, and gender<br>(systolic and/or diastolic) | ≥ 95th percentile adjusted for age, height, and gender (systolic and/or diastolic) | Life-threatening consequences<br>(eg, malignant hypertension)<br>OR Hospitalization indicated<br>(other than emergency room<br>visit) |
| Hypotension | NA | Symptomatic, corrected with oral fluid replacement | Symptomatic, IV fluids indicated | Shock requiring use of vasopressors or mechanical assistance to maintain blood pressure |
| Pericardial Effusion | Asymptomatic, small effusion requiring no intervention | Asymptomatic, moderate or larger effusion requiring no intervention | Effusion with non-life-<br>threatening physiologic<br>consequences OR Effusion<br>with nonurgent intervention<br>indicated | Life-threatening consequences<br>(eg, tamponade) OR Urgent<br>intervention indicated |

| | CARDIOVASCULAR | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Prolonged PR Interval | PR interval 0.21 to 0.25 sec | PR interval > 0.25 sec | Type II 2nd degree AV<br>block OR Ventricular pause<br>> 3.0 sec | Complete AV block |
| Pediatric ≤ 16 Years | 1st degree AV block<br>(PR > normal for age and rate) | Type I 2nd degree AV block | Type II 2nd degree AV block | Complete AV block |
| Prolonged QTc | Asymptomatic, QTc interval 0.45 to 0.47 sec OR Increase interval < 0.03 sec above baseline | Asymptomatic, QTc interval 0.48 to 0.49 sec OR Increase in interval 0.03 to 0.05 sec above baseline | Asymptomatic, QTc interval ≥ 0.50 sec OR Increase in interval ≥ 0.06 sec above baseline | Life-threatening consequences, eg, Torsade de pointes or other associated serious ventricular dysrhythmia |
| Pediatric ≤ 16 Years | Asymptomatic, QTc interval 0.450 to 0.464 sec | Asymptomatic, QTc interval 0.465 to 0.479 sec | Asymptomatic, QTc interval ≥ 0.480 sec | Life-threatening consequences, eg, Torsade de pointes or other associated serious ventricular dysrhythmia |
| Thrombosis/Embolism | NA | Deep vein thrombosis AND<br>No intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Deep vein thrombosis AND<br>Intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Embolic event (eg, pulmonary embolism, life-threatening thrombus) |
| Vasovagal Episode (associated with a procedure of any kind) | Present without loss of consciousness | Present with transient loss of consciousness | NA | NA |
| Ventricular Dysfunction<br>(congestive heart failure,<br>CHF) | NA | Asymptomatic diagnostic finding AND intervention indicated | New onset with symptoms<br>OR Worsening symptomatic<br>CHF | Life-threatening CHF |

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bronchospasm (acute) | FEV1 or peak flow reduced to 70% to 80% | FEV1 or peak flow 50% to 69% | FEV1 or peak flow 25% to 49% | Cyanosis OR FEV1 or peak flow < 25% OR Intubation |
| Dyspnea or Respiratory<br>Distress | Dyspnea on exertion with no or minimal interference with usual social & functional activities | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities | Dyspnea at rest causing inability to perform usual social & functional activities | Respiratory failure with ventilatory support indicated |
| Pediatric < 14 Years | Wheezing OR minimal increase in respiratory rate for age | Nasal flaring OR Intercostal retractions OR Pulse oximetry 90% to 95% | Dyspnea at rest causing inability to perform usual social & functional activities OR Pulse oximetry < 90% | Respiratory failure with ventilatory support indicated |

| OCULAR/VISUAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Uveitis | Asymptomatic but detectable on exam | Symptomatic anterior uveitis OR Medical intervention indicated | Posterior or pan-uveitis OR<br>Operative intervention<br>indicated | Disabling visual loss in affected eye(s) |
| Visual Changes (from baseline) | Visual changes causing no or minimal interference with usual social & functional activities | Visual changes causing greater than minimal interference with usual social & functional activities | Visual changes causing inability to perform usual social & functional activities | Disabling visual loss in affected eye(s) |

| | SKIN | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alopecia | Thinning detectable by study participant or caregiver (for disabled adults) | Thinning or patchy hair loss detectable by health care provider | Complete hair loss | NA |
| Cutaneous Reaction – Rash | Localized macular rash | Diffuse macular,<br>maculopapular, or<br>morbilliform rash OR Target<br>lesions | Diffuse macular,<br>maculopapular, or morbilliform<br>rash with vesicles or limited<br>number of bullae OR<br>Superficial ulcerations of<br>mucous membrane limited to<br>one site | Extensive or generalized<br>bullous lesions OR<br>Stevens-Johnson syndrome<br>OR Ulceration of mucous<br>membrane involving two<br>or more distinct mucosal<br>sites OR Toxic epidermal<br>necrolysis (TEN) |
| Hyperpigmentation | Slight or localized | Marked or generalized | NA | NA |
| Hypopigmentation | Slight or localized | Marked or generalized | NA | NA |
| Pruritis (itching – no skin lesions) (See also Injection Site Reactions: Pruritis associated with injection) | Itching causing no or<br>minimal interference with<br>usual social & functional<br>activities | Itching causing greater than minimal interference with usual social & functional activities | Itching causing inability to perform usual social & functional activities | NA |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite associated with decreased oral intake without significant weight loss | Loss of appetite associated with significant weight loss | Life-threatening consequences<br>OR Aggressive intervention<br>indicated [eg, tube feeding or<br>total parenteral nutrition] |
| Ascites | Asymptomatic | Symptomatic AND Intervention indicated (eg, diuretics or therapeutic paracentesis) | Symptomatic despite intervention | Life-threatening consequences |
| Cholecystitis | NA | Symptomatic AND Medical intervention indicated | Radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences (eg, sepsis or perforation) |
| Constipation | NA | Persistent constipation requiring regular use of dietary modifications, laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening consequences (eg, obstruction) |
| Diarrhea | | | | |
| Adult and Pediatric<br>≥1 Year | Transient or intermittent episodes of unformed stools OR Increase of ≤ 3 stools over baseline/24 hr | Persistent episodes of unformed to watery stools OR Increase of 4–6 stools over baseline per 24 hrs. | Bloody diarrhea OR Increase<br>of ≥ 7 stools per 24-hour<br>period OR IV fluid<br>replacement indicated | Life-threatening consequences (eg, hypotensive shock) |
| Pediatric < 1 Year | Liquid stools (more unformed than usual) but usual number of stools | Liquid stools with increased<br>number of stools OR Mild<br>dehydration | Liquid stools with moderate dehydration | Liquid stools resulting in<br>severe dehydration with<br>aggressive rehydration<br>indicated OR Hypotensive<br>shock |
| Dysphagia-Odynophagia | Symptomatic but able to eat usual diet | Symptoms causing altered dietary intake without medical intervention indicated | Symptoms causing severely altered dietary intake with medical intervention indicated | Life-threatening reduction in oral intake |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucositis/Stomatitis<br>(clinical exam) See also Proctitis,<br>Dysphagia-Odynophagia | Erythema of the mucosa | Patchy pseudomembranes or ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Tissue necrosis OR Diffuse<br>spontaneous mucosal bleeding<br>OR Life-threatening<br>consequences (eg, aspiration,<br>choking) |
| Nausea | Transient (< 24 hours) or intermittent nausea with no or minimal interference with oral intake | Persistent nausea resulting in decreased oral intake for 24–48 hours | Persistent nausea resulting in minimal oral intake for > 48 hours OR Aggressive rehydration indicated (eg, IV fluids) | Life-threatening consequences (eg, hypotensive shock) |
| Pancreatitis | NA | Symptomatic AND<br>Hospitalization not indicated<br>(other than ER visit) | Symptomatic AND<br>Hospitalization indicated<br>(other than ER visit) | Life-threatening consequences<br>(eg, sepsis, circulatory failure,<br>hemorrhage) |
| Proctitis (functional-<br>symptomatic) Also see Mucositis/<br>Stomatitis for Clinical<br>Exam | Rectal discomfort AND No intervention indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social/ functional activities OR Operative intervention indicated | Life-threatening consequences (eg, perforation) |
| Vomiting | Transient or intermittent vomiting with no or minimal interference with oral intake | Frequent episodes of vomiting with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated | Life-threatening consequences (eg, hypotensive shock) |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alteration in Personality-<br>Behavior or in Mood (eg,<br>agitation, anxiety,<br>depression, mania,<br>psychosis) | Alteration causing no or minimal interference with usual social & functional activities | Alteration causing greater than minimal interference with usual social & functional activities | Alteration causing inability to perform usual social & functional activities | Behavior potentially harmful<br>to self or others (eg,<br>suicidal/homicidal ideation or<br>attempt, acute psychosis) OR<br>Causing inability to perform<br>basic self-care functions |
| Altered Mental Status For Dementia, see Cognitive and Behavioral/Attentional Disturbance (including dementia and ADD) | Changes causing no or minimal interference with usual social & functional activities | Mild lethargy or somnolence causing greater than minimal interference with usual social & functional activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR obtundation, OR coma |
| Ataxia | Asymptomatic ataxia detectable on exam OR Minimal ataxia causing no or minimal interference with usual social & functional activities | Symptomatic ataxia causing greater than minimal interference with usual social & functional activities | Symptomatic ataxia causing inability to perform usual social & functional activities | Disabling ataxia causing inability to perform basic self-care functions |
| Cognitive and Behavioral/Attentional Disturbance (including dementia and Attention Deficit Disorder) | Disability causing no or<br>minimal interference with<br>usual social & functional<br>activities OR Specialized<br>resources not indicated | Disability causing greater than minimal interference with usual social & functional activities OR Specialized resources on part-time basis indicated | Disability causing inability to perform usual social & functional activities OR Specialized resources on a full-time basis indicated | Disability causing inability to perform basic self-care functions OR Institutionalization indicated |
| CNS Ischemia (acute) | NA | NA | Transient ischemic attack | Cerebral vascular accident (CVA, stroke) with neurological deficit |

| | | NEUROLOGICAL | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Developmental delay – Pediatric ≤ 16 Years | Mild developmental delay,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate<br>for the setting | Moderate developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Severe developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Developmental regression,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate for<br>the setting |
| Headache | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated (other than ER visit) OR Headache with significant impairment of alertness or other neurologic function |
| Insomnia | NA | Difficulty sleeping causing greater than minimal interference with usual social/functional activities | Difficulty sleeping causing inability to perform usual social & functional activities | Disabling insomnia causing inability to perform basic self-care functions |
| Neuromuscular Weakness (including myopathy & neuropathy) | Asymptomatic with decreased strength on exam OR Minimal muscle weakness causing no or minimal interference with usual social & functional activities | Muscle weakness causing greater than minimal interference with usual social & functional activities | Muscle weakness causing inability to perform usual social & functional activities | Disabling muscle weakness causing inability to perform basic self-care functions OR Respiratory muscle weakness impairing ventilation |
| Neurosensory Alteration<br>(including paresthesia and<br>painful neuropathy) | Asymptomatic with sensory alteration on exam or minimal paresthesia causing no or minimal interference with usual social & functional activities | Sensory alteration or<br>paresthesia causing greater<br>than minimal interference with<br>usual social & functional<br>activities | Sensory alteration or<br>paresthesia causing inability to<br>perform usual social &<br>functional activities | Disabling sensory alteration or<br>paresthesia causing inability to<br>perform basic self-care<br>functions |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 Grade 2 Grade 3 Grade 4 | | | |
| Seizure: (new onset) | NA | 1 seizure | 2–4 seizures | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure: (pre-existing) For Worsening of Existing Epilepsy the Grades Should Be Based on an Increase from Previous Level of Control to Any of These Levels | NA | Increased frequency of pre-<br>existing seizures (non-<br>repetitive) without change in<br>seizure character OR<br>infrequent breakthrough<br>seizures while on stable meds<br>in a previously controlled<br>seizure disorder | Change in seizure character<br>from baseline either in<br>duration or quality (eg,<br>severity or focality) | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure - Pediatric < 18 Years | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>< 5 minutes with < 24 hours<br>post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting 5–20<br>minutes with<br>< 24 hours post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>> 20 minutes | Seizure, generalized onset<br>with or without secondary<br>generalization, requiring<br>intubation and sedation |
| Syncope (not associated with a procedure) | NA | Present | NA | NA |
| Vertigo | Vertigo causing no or<br>minimal interference with<br>usual social & functional<br>activities | Vertigo causing greater than minimal interference with usual social & functional activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo causing inability to perform basic self-care functions |

| | MUSCULOSKELETAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia See also Arthritis | Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain causing inability to perform basic self-care functions |
| Arthritis See also Arthralgia | Stiffness or joint swelling causing no or minimal interference with usual social & functional activities | Stiffness or joint swelling causing greater than minimal interference with usual social & functional activities | Stiffness or joint swelling causing inability to perform usual social & functional activities | Disabling joint stiffness or<br>swelling causing inability to<br>perform basic self-care<br>functions |
| Bone Mineral Loss | BMD t-score or z-score<br>-2.5 to -1.0 | BMD t-score or z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Pediatric < 21 Years | BMD z-score<br>-2.5 to -1.0 | BMD z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Myalgia<br>(non-injection site) | Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain causing inability to perform basic self-care functions |
| Osteonecrosis | NA | Asymptomatic with radiographic findings AND No operative intervention indicated | Symptomatic bone pain with radiographic findings OR Operative intervention indicated | Disabling bone pain with radiographic findings causing inability to perform basic self-care functions |

| | SYSTEMIC | | | |
|---|---|---|---|---|
| | Grade 1 Grade 2 Grade 3 Grade 4 | | | |
| Acute Systemic Allergic<br>Reaction | (wheals) with no medical intervention indicated OR Mild angioedema with no medical intervention indicated | | Generalized urticaria OR<br>Angioedema with medical<br>intervention indicated OR<br>Symptomatic mild<br>bronchospasm | Acute anaphylaxis OR Life-<br>threatening bronchospasm OR<br>laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | imal interference with minimal interference with usual social & functional social & functional activities | | NA |
| Fatigue<br>Malaise | Symptoms causing no or minimal interference with usual social & functional activities | mal interference with social & functional social & functional | | Incapacitating fatigue/malaise symptoms causing inability to perform basic self-care functions |
| Fever (nonaxillary) | 37.7°C to 38.6°C<br>99.8°F to 101.5°F | 38.7°C to 39.3°C<br>101.6°F to 102.8°F | 39.4°C to 40.5°C<br>102.9°F to 104.9°F | > 40.5°C<br>> 104.9°F |
| Pain- Indicate Body Site See also Injection Site Pain, Headache, Arthralgia, and Myalgia | Pain causing no or<br>minimal interference with<br>usual social & functional<br>activities | Pain causing greater than minimal interference with usual social & functional activities | Pain causing inability to perform usual social & functional activities | Disabling pain causing inability to perform basic self-care functions OR Hospitalization (other than ER visit) indicated |
| Unintentional Weight<br>Loss | NA | 5% to 9% loss in body weight from baseline | 10% to 19% loss in body weight from baseline | ≥ 20% loss in body weight<br>from baseline OR Aggressive<br>intervention indicated [eg,<br>tube feeding or total parenteral<br>nutrition] |

| | INJECTION SITE REACTION | | | |
|---|---|---|---|---|
| | Grade 3 | Grade 4 | | |
| Injection Site Pain (pain without touching) Or Tenderness (pain when area is touched) | Pain/tenderness causing no or minimal limitation of use of limb | Pain/tenderness limiting use of limb OR Pain/tenderness causing greater than minimal interference with usual social & functional activities | Pain/tenderness causing inability to perform usual social & functional activities | Pain/tenderness causing inability<br>to perform basic self-care<br>function OR Hospitalization<br>(other than ER visit) indicated<br>for management of<br>pain/tenderness |
| Injection Site Reaction (Localized), > 15 Years | Erythema OR Induration<br>of $5 \times 5$ cm to $9 \times 9$ cm (or<br>$25-81 \times \text{cm}^2$ ) | Erythema OR Induration OR<br>Edema > 9 cm any diameter<br>(or > 81 cm <sup>2</sup> ) | Ulceration OR Secondary<br>infection OR Phlebitis OR<br>Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pediatric ≤ 15 Years | Erythema OR Induration<br>OR Edema present but<br>≤ 2.5 cm diameter | Erythema OR Induration<br>OR Edema > 2.5 cm<br>diameter but < 50% surface<br>area of the extremity<br>segment (eg, upper<br>arm/thigh) | Erythema OR Induration OR Edema involving ≥ 50% surface area of the extremity segment (eg, upper arm/thigh) OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pruritis Associated with Injection See also Skin: Pruritis (itching—no skin lesions) | Itching localized to injection<br>site AND Relieved<br>spontaneously or with<br>< 48 h treatment | Itching beyond the injection site but not generalized OR Itching localized to injection site requiring ≥ 48 h treatment | Generalized itching causing inability to perform usual social & functional activities | NA |

| | ENDOCRINE/METABOLIC | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Lipodystrophy (eg, back of neck, breasts, abdomen) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious changes on casual visual inspection | NA |
| Diabetes Mellitus | NA | New onset without need to initiate medication OR Modification of current meds to regain glucose control | New onset with initiation of indicated med OR Diabetes uncontrolled despite treatment modification | Life-threatening consequences<br>(eg, ketoacidosis,<br>hyperosmolar non-ketotic<br>coma) |
| Gynecomastia | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |
| Hyperthyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, thyroid storm) |
| Hypothyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, myxedema coma) |
| Lipoatrophy (eg, fat loss from the face, extremities, buttocks) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |

| | GENITOURINARY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Intermenstrual Bleeding (IMB) | Spotting observed by participant OR Minimal blood observed during clinical or colposcopic exam | Intermenstrual bleeding not greater in duration or amount than usual menstrual cycle | Intermenstrual bleeding greater in duration or amount than usual menstrual cycle | Hemorrhage with life-<br>threatening hypotension OR<br>Operative intervention<br>indicated |
| Urinary Tract obstruction (eg, stone) | NA | Signs or symptoms of urinary tract obstruction without hydronephrosis or renal dysfunction | Signs or symptoms of urinary tract obstruction with hydronephrosis or renal dysfunction | Obstruction causing life-<br>threatening consequences |

| INFECTION | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Infection (any other than HIV infection) | Localized, no systemic antiµbial treatment indicated AND Symptoms causing no or minimal interference with usual social & functional activities | Systemic antiµbial treatment indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Systemic antiµbial treatment indicated AND Symptoms causing inability to perform usual social & functional activities OR Operative intervention (other than simple incision and drainage) indicated | Life-threatening consequences (eg, septic shock) |

Basic Self-care Functions: Activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding.

Usual Social & Functional Activities: Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, pursuing a hobby, etc

# Appendix 4. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

# 1) Background

Non-clinical toxicity studies of sofosbuvir and ledipasvir demonstrated no adverse effect on embryo-fetal development. However, there are no clinical studies of sofosbuvir or ledipasvir in pregnant women. Please refer to the latest version of the investigator's brochure for additional information

2) Definition of Female of Childbearing Potential and Contraceptive Requirements for Female Subjects (and their male partners)

Women > 54 years of age with cessation for  $\geq$  12 months of previously occurring menses, or women of any age who have had a hysterectomy, or have had both ovaries removed, or have had medically documented ovarian failure will be considered to be of non-childbearing potential.

Women  $\leq$  54 years of age (including those with amenorrhea of any duration) who have not had a hysterectomy, and have not had both ovaries removed, and have not had medically documented ovarian failure will be considered to be of childbearing potential.

Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on the Baseline/Day 1 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Baseline/Day 1 until 30 days after last dose of study drug.

• <u>Complete</u> abstinence from intercourse. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

#### Or

| • | Consistent and correct use of 1 of the following methods of birth control listed below, in |
|---|---|
| | addition to a male partner who correctly uses a condom, from the date of Screening until |
| | 30 days after last dose of study drug: |

| <br>intrauterine device (IUD) with a failure rate of < 1% per year |
|-----------------------------------------------------------------------------|
| <br>female barrier method: cervical cap or diaphragm with spermicidal agent |
| <br>tubal sterilization |
| <br>vasectomy in male partner |
| <br>hormone-containing contraceptive: |

- injectable progesterone
- oral contraceptives (either combined or progesterone only)
- contraceptive vaginal ring
- transdermal contraceptive patch
- 3) Contraceptive Requirements for Male Subjects (and their female partners)

All male study participants must agree to consistently and correctly use a condom from the date of Screening until 90 days after the last dose of study drug. If their female partner is of child bearing potential (as defined above), their female partner must use 1 of the methods of birth control listed above from the date of Screening until 90 days after the last dose of study drug.

Male subjects must agree to refrain from sperm donation for at least 90 days after the last dose of study drug.

## 4) Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they (or their partner) become pregnant at any time during the study, or if they become pregnant within 30 days (90 days for partners of male subjects) of last study drug dose. Subjects who become pregnant or who suspect that they are pregnant must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant must report the information to the investigator.

Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 7.7.2.1.

# Appendix 5. Calculation of Historical Control SVR12 for Treatment-naïve Korean Subjects and for Treatment-naïve Chinese Subjects with Chronic GT-1 HCV Infection

This section details the calculation for the historical control SVR12 rates for treatment-naïve Korean subjects and for treatment-naïve Chinese subjects with chronic GT-1 HCV infection.

The historical control calculation for Korea assumes that of the treatment-naïve subjects with HCV GT-1 infection to be enrolled in Korea, approximately 60% will have 'Uncomplicated Infection', ~30% will be 'Elderly', and ~10% will be 'Cirrhotic'. Based on discussions with clinical investigators in these countries, these assumptions ensure a conservative estimation of the historical SVR rate following Peg-IFN $\alpha$ +RBV in the respective populations. The references used for the calculation of the historical control rates are provided in Appendix Table 2 below.

For Korea, the SVR rates among each of the three patient populations are calculated according to the reference studies (Appendix Table 2). The overall historical SVR rate is subsequently calculated as the weighted average of the population-specific rates, with the weight being the expected percentages of patients in each population. With these assumptions in mind and using the referenced literature, the adjusted historical SVR control rate for the populations in Korea are calculated as follows:

Appendix Table 1. SVR rates following Peg-IFNα+RBV in Treatment-Naïve Korean Subjects with GT-1 HCV Infection

| Country | Uncomplicated<br>Infection | Elderly | Cirrhotic | Weighted Average |
|---|---|---|---|---|
| Korea | 62.7% | 30.8% | 24% | 62.7% * 0.6 + 30.8% * 0.3 + 24% *0.1= 49% |

Therefore, a null adjusted historical SVR rate for this study is 49% following estimation of the SVR rate for Korea.

For China, the historical control rate has been calculated according to the reference studies in Appendix Table 3. SVR rates are not reported separately for elderly patients or those with cirrhosis in these references. Consequently, the calculated historical SVR rate of 57% has not been adjusted by different population.

Appendix Table 2. Literature References for Historical Control Rate Calculations in Korea

| SVR | Rates in I | Korea | |
|---|---|---|---|
| Population | SVR% | SVR n/N | Reference |
| | 80.8 | 21/26 | {24236} |
| | 54.7 | 58/106 | {24236} |
| CT 1 Treatment Navies (Day IEN/DDV 40 Weeks) | 62.7 | 341/543 | {26807} |
| GT-1 Treatment Naïve (Peg-IFN/RBV 48 Weeks) | 62.2 | 158/254 | {26389} |
| | 64.2 | 104/162 | {26389} |
| | 66.0 | 31/47 | {26390} |
| Overall SVR Rate | 62.7% | | |
| SVR Rat | es in Kore | a Elderly | |
| Population | SVR% | SVR n/N | Reference |
| GT-1 Treatment Naïve (Peg-IFN/RBV 48 weeks) | 30.8 | 4/13 | {26390} |
| Overall SVR Rate | | | 30.8% |
| SVR Rates in Korea Cirrhotics | | | |
| Population | SVR% | SVR n/N | Reference |
| GT-1 Treatment Naïve (Peg-IFN/RBV 48 weeks) | 24.0 | 12/50 | {24405} |
| Overall SVR Rate | | | 24.0% |

**Appendix Table 3.** Literature References for Historical Control Rate Calculations in China

| SVR Rates in China | | | |
|---|---|---|---|
| Population SVR % SVR n/N Reference | | | |
| GT-1 Treatment Naïve (Peg-IFN/RBV 48 weeks) | 70.3 | 102/145 | {24797} |
| | 43.9 | 18/41 | {13261} |
| | 46.0 | 58/126 | {24391} |
| Overall SVR Rate | | (102+18+ | <del>-58)</del> / (145+41+126) = 57% |